

# COVID-19: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD CROSSOVER STUDY TO ESTIMATE THE EFFECT OF ITRACONAZOLE ON THE PHARMACOKINETICS OF PF-07321332/RITONAVIR IN HEALTHY PARTICIPANTS

**Study Intervention Number:** PF-07321332

**Study Intervention Name:** N/A

**US IND Number:** 153517

**EudraCT Number:** 2021-003308-42

ClinicalTrials.gov ID: N/A

**Protocol Number:** C4671015

Phase:

**Brief Title:** A Phase 1 Study to Estimate the Effect of Itraconazole on the PK of PF-07321332/Ritonavir in Healthy Participants

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# **Document History**

| Document | Version Date |
|-------------------|--------------|
| Amendment 1 | 02 July 2021 |
| Original protocol | 15 June 2021 |

This amendment incorporates all revisions to date, including amendments made at the request of country health authorities and IRBs/ECs and any global protocol administrative clarification letter.

# **Protocol Amendment Summary of Changes Table**

# **Amendment 1 (02-July-2021)**

**Overall Rationale for the Amendment:** This study is being amended to reflect changes in response to comments from Competent Authority/Ethics Committee. Detailed changes are summarized below in a tabular form.

| Section # and<br>Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Section 1.3 Schedule of | Remove "Pharmacogenomic blood sampling" | • Updates made to reflect the current design of the study. |
| Activities | • CCI | • CCI |
| Section 5.2<br>Exclusion Criteria | Updated the exclusion criterion #14 to "AST or ALT level > 1.0 × ULN". | Participants should be excluded if their AST or ALT levels are greater than (>) the ULN. |
| Section 7.1.2<br>Potential Cases of<br>Acute Kidney Injury | Specify that the described increase of SCr should trigger a halt/stopping of dosing. | Updates made to respond to comments from Competent Authority/Ethics Committee. |
| Section 7.1.3 | Added Section 7.1.3 "Stopping Rules" | Updates made to respond to comments from Competent Authority/Ethics Committee. |

| Section # and<br>Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Original Section<br>8.5.3<br>Pharmacogenomic<br>Sample | Removed Section 8.5.3<br>Pharmacogenomic Sample | Updates made to reflect the current design of the study. |
| CCI | • CCI | . CCI |
| Section 10.6<br>Appendix 6. | Specify that the described liver function abnormalities should trigger a halt/stopping of dosing. | Updates made to respond to comments from Competent Authority/Ethics Committee. |
| | Minor editorial changes throughout. | |

# **TABLE OF CONTENTS**

| LIST OF TABLES | 8 |
|-----------------------------------------------------------|----|
| 1. PROTOCOL SUMMARY | 9 |
| 1.1. Synopsis | 9 |
| 1.2. Schema | 13 |
| 1.3. Schedule of Activities | 14 |
| 2. INTRODUCTION | 18 |
| 2.1. Study Rationale | 18 |
| 2.2. Background | 18 |
| 2.2.1. Nonclinical Pharmacology | 18 |
| 2.2.2. Nonclinical Pharmacokinetics and Metabolism | 18 |
| 2.2.3. Nonclinical Safety | 19 |
| 2.2.4. Clinical Overview | |
| 2.2.4.1. Safety Overview | 20 |
| 2.2.4.2. Summary of PF-07321332 Pharmacokinetics in Human | 20 |
| 2.3. Benefit/Risk Assessment | 21 |
| 2.3.1. Risk Assessment | 22 |
| 2.3.2. Benefit Assessment | 25 |
| 2.3.3. Overall Benefit/Risk Conclusion | 25 |
| 3. OBJECTIVES AND ENDPOINTS | 25 |
| 4. STUDY DESIGN | 25 |
| 4.1. Overall Design. | 25 |
| 4.2. Scientific Rationale for Study Design | 26 |
| 4.2.1. Choice of Contraception/Barrier Requirements | 27 |
| 4.2.2. Collection of Retained Research Samples | 27 |
| 4.3. Justification for Dose | 27 |
| 4.4. End of Study Definition | 28 |
| 5. STUDY POPULATION | 28 |
| 5.1. Inclusion Criteria | 28 |
| 5.2. Exclusion Criteria | 29 |
| 5.3. Lifestyle Considerations | 31 |

| 5.3.1. Meals and Dietary Restrictions | 31 |
|---|---|
| 5.3.2. Caffeine, Alcohol, and Tobacco | 32 |
| 5.3.3. Activity | 33 |
| 5.3.4. Contraception | 33 |
| 5.4. Screen Failures | 33 |
| 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY | 33 |
| 6.1. Study Intervention(s) Administered | 33 |
| 6.1.1. Administration | 34 |
| 6.2. Preparation, Handling, Storage, and Accountability | 35 |
| 6.2.1. Preparation and Dispensing | 36 |
| 6.3. Measures to Minimize Bias: Randomization and Blinding | 36 |
| 6.3.1. Allocation to Study Intervention | 36 |
| 6.4. Study Intervention Compliance | 37 |
| 6.5. Dose Modification | 37 |
| 6.6. Continued Access to Study Intervention After the End of the Study | 37 |
| 6.7. Treatment of Overdose | 37 |
| 6.8. Concomitant Therapy | 37 |
| 6.8.1. Rescue Medicine | 38 |
| 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 38 |
| 7.1. Discontinuation of Study Intervention | 38 |
| 7.1.1. ECG Changes | 38 |
| 7.1.2. Potential Cases of Acute Kidney Injury | 39 |
| 7.1.3. Stopping Rules | |
| 7.2. Participant Discontinuation/Withdrawal From the Study | 40 |
| 7.2.1. Withdrawal of Consent | 40 |
| 7.3. Lost to Follow up | 41 |
| 8. STUDY ASSESSMENTS AND PROCEDURES | 41 |
| 8.1. Efficacy Assessments | 42 |
| 8.2. Safety Assessments | 42 |
| 8.2.1. Physical Examinations | |
| 8.2.2. Vital Signs | 43 |

| 8.2.2.1. Respiratory Rate | 43 |
|---|---|
| 8.2.2.2. Temperature | 44 |
| 8.2.3. Electrocardiograms | 44 |
| 8.2.4. Clinical Safety Laboratory Assessments | 44 |
| 8.2.5. COVID-19 Specific Assessments | 45 |
| 8.2.6. Pregnancy Testing | 45 |
| 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting | 45 |
| 8.3.1. Time Period and Frequency for Collecting AE and SAE Information | 46 |
| 8.3.1.1. Reporting SAEs to Pfizer Safety | 46 |
| 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF | 47 |
| 8.3.2. Method of Detecting AEs and SAEs | 47 |
| 8.3.3. Follow-Up of AEs and SAEs | 47 |
| 8.3.4. Regulatory Reporting Requirements for SAEs | 47 |
| 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure | 48 |
| 8.3.5.1. Exposure During Pregnancy | 48 |
| 8.3.5.2. Exposure During Breastfeeding | 50 |
| 8.3.5.3. Occupational Exposure | 50 |
| 8.3.6. Cardiovascular and Death Events | 50 |
| 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs | 50 |
| 8.3.8. Adverse Events of Special Interest | 50 |
| 8.3.8.1. Lack of Efficacy | 51 |
| 8.3.9. Medical Device Deficiencies | 51 |
| 8.3.10. Medication Errors | 51 |
| 8.4. Pharmacokinetics | 52 |
| 8.4.1. Plasma for Analysis of PF-07321332 CCI | 52 |
| 8.5. Genetics | 53 |
| 8.5.1. Specified Genetics | 53 |
| CCI | |
| 8.6. Biomarkers | 53 |
| 8.6.1. Specified Gene Expression (RNA) Research | 53 |

| 8.6.2. Specified Protein Research | 53 |
|---|---|
| 8.6.3. Specified Metabolomic Research | 53 |
| CCI | |
| 8.7. Immunogenicity Assessments | 54 |
| 8.8. Health Economics | 54 |
| 9. STATISTICAL CONSIDERATIONS | 54 |
| 9.1. Statistical Hypotheses | 54 |
| 9.2. Analysis Sets | 54 |
| 9.3. Statistical Analyses | 55 |
| 9.3.1. Pharmacokinetic Analyses | 55 |
| 9.3.1.1. Derivation of Pharmacokinetic Parameters | 55 |
| 9.3.2. Statistical Methods for PK Data | 55 |
| 9.3.3. Other Safety Analyses | 56 |
| CCI | |
| 9.4. Interim Analyses | 56 |
| 9.5. Sample Size Determination | 56 |
| 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 58 |
| 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 58 |
| 10.1.1. Regulatory and Ethical Considerations | 58 |
| 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 58 |
| 10.1.2. Informed Consent Process | 59 |
| 10.1.3. Data Protection | 60 |
| 10.1.4. Committees Structure | 60 |
| 10.1.4.1. Data Monitoring Committee | 60 |
| 10.1.5. Dissemination of Clinical Study Data | 60 |
| 10.1.6. Data Quality Assurance | 61 |
| 10.1.7. Source Documents | 62 |
| 10.1.8. Study and Site Start and Closure | 63 |
| 10.1.9. Publication Policy | 64 |
| 10.1.10. Sponsor's Qualified Medical Personnel | 64 |

| 10.2. | Appendix 2: Clinical Laboratory Tests | 66 |
|---|---|---|
| | Appendix 3: Adverse Events: Definitions and Procedures for Recording, valuating, Follow-Up, and Reporting | 67 |
| | 10.3.1. Definition of AE | 67 |
| | 10.3.2. Definition of an SAE | 68 |
| | 10.3.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period | 69 |
| | 10.3.4. Reporting of SAEs | 73 |
| 10.4. | Appendix 4: Contraceptive and Barrier Guidance | 74 |
| | 10.4.1. Male Participant Reproductive Inclusion Criteria | 74 |
| | 10.4.2. Female Participant Reproductive Inclusion Criteria | 74 |
| | 10.4.3. Woman of Childbearing Potential | 75 |
| | 10.4.4. Contraception Methods | 76 |
| CCI | | |
| 10.6. | Appendix 6: Liver Safety: Suggested Actions and Follow-Up Assessments | 78 |
| 10.7. | Appendix 7: ECG Findings of Potential Clinical Concern | 80 |
| 10.8. | Appendix 8: Abbreviations | 82 |
| 11. REFER | RENCES | 86 |
| | LIST OF TABLES | |
| Table 1. | Protocol-Required Safety Laboratory Assessments | 66 |

#### 1. PROTOCOL SUMMARY

# 1.1. Synopsis

**Brief Title:** A Phase 1 Study to Estimate the Effect of Itraconazole on the PK of PF-07321332/Ritonavir in Healthy Participants

#### Rationale

PF-07321332 is a potent and selective inhibitor of the SARS-CoV-2 3CL protease that is currently being developed as an oral treatment of COVID-19. Ritonavir is a strong CYP3A4 inhibitor being used to inhibit the metabolism of PF-07321332 in order to increase plasma concentrations of PF-07321332 to values that are anticipated to be efficacious.

In vitro and in vivo metabolite profiling suggests that the primary clearance mechanism for PF-07321332 is CYP3A4 mediated oxidation. In a reaction phenotyping study using human liver microsomes in the presence of selective CYP inhibitors, CYP3A4 was predicted to be the major contributor ( $f_m = 0.99$ ) to the in vitro oxidative metabolism of PF-07321332. As such, in the FIH Study, C4671001, the CYP3A4 inhibitor ritonavir was used to enhance the exposure of PF-07321332 in order to achieve plasma levels that are anticipated to be efficacious. Preliminary PK data following multiple oral administrations of PF-07321332/ritonavir at doses of 75/100 mg to 500/100 mg q12h suggest that the renal pathway may also play a significant role in PF-07321332 excretion when co-administered with ritonavir (32.5% to 64.6% of the drug excreted unchanged in urine across doses at steady-state). Ritonavir is extensively metabolized, primarily by CYP3A4. Mechanistically, inhibition of CYP3A4 could further decrease the metabolism of PF-07321332 and ritonavir, and thereby increase circulating exposures.

The purpose of this study is to estimate the effect of a strong inhibitor of CYP3A4 on the PK of PF-07321332/ritonavir in healthy participants.

# **Objectives and Endpoints**

| Primary Objective: | Primary Endpoint: |
|---|---|
| To estimate the effect of multiple doses of itraconazole on the PK of PF-07321332 following multiple doses of PF-07321332/ritonavir | PF-07321332 plasma PK parameters: C <sub>max</sub> and AUC <sub>tau</sub> with itraconazole (test) versus without itraconazole (reference) |
| Secondary Objective: | Secondary Endpoints: |
| <ul> <li>To evaluate the safety and tolerability of PF-07321332/ritonavir in healthy participants in the absence and presence of multiple doses of itraconazole</li> <li>To characterize the PK of PF-07321332 following multiple doses when PF-07321332/ritonavir is administered alone or with itraconazole in healthy participants.</li> </ul> | <ul> <li>Assessment of TEAEs, clinical laboratory abnormalities, vital signs, physical exam, and 12-lead ECGs</li> <li>PF-07321332 plasma PK parameters: T<sub>max</sub>, t<sub>1/2</sub>, AUC<sub>last</sub>, CL/F, and V<sub>z</sub>/F for PF-07321332 with and without coadministration of itraconazole.</li> </ul> |
| CCI | |

# **Overall Design**

#### **Brief Summary**

This is a Phase 1, open-label, 2-period, fixed sequence crossover study to estimate the effect of the strong CYP3A4 inhibitor, itraconazole, on the PK of PF-07321332 and ritonavir in healthy participants. The study will consist of 2 treatments: multiple oral doses of 300 mg PF-07321332/100 mg ritonavir alone and multiple oral doses of 300 mg PF-07321332/100 mg ritonavir in combination with itraconazole. A total of approximately 12 healthy male and/or female participants will be enrolled into the study to ensure at least 9 participants will complete the study. The treatment will consist of a single fixed sequence. Participants who discontinue from the study for non-safety reasons may be replaced at the sponsor's discretion in collaboration with the Investigator.

Healthy participants will be screened to determine eligibility within 28 days prior to study treatment. Medical history and results of physical examination, physical measurements, vital signs, 12-lead ECGs, and clinical laboratory evaluations will determine eligibility. Participants will report to the CRU on Day -1 and will be required to stay in the CRU for 14 days and 13 nights.

In Period 1, each enrolled participant will receive 300 mg PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses, from Day 1 morning to Day 3 morning. Serial PK samples will be collected up to 48 hours post the 5<sup>th</sup> dose on Day 3 to establish baseline

exposure of PF-07321332. PK samples will also be collected predose the morning and evening doses of PF-07321332/ritonavir on Day 2 to confirm steady state.

Period 2 will begin on Study Day 5 (referred to as Period 2, Day 1). Participants will receive 200 mg itraconazole, administered orally, QD, on Period 2, Days 1 through 8, inclusive. On Days 4, 5, and 6, participants will receive 300 mg PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses, from Period 2, Day 4 morning to Day 6 morning. Following the final administration of PF-07321332/ritonavir on the morning of Day 6, participants will undergo serial PK sampling up to 72 hours post the last dose. PK samples will also be collected predose the morning and evening doses of PF-07321332/ritonavir on Day 5 to confirm steady state. Participants will be discharged from the CRU on Period 2, Day 9 following completion of all assessments.

If a participant has any clinically significant, study related abnormalities at the conclusion of a scheduled inpatient portion of the study, the Pfizer medical monitor (or designated representative) should be notified and the participant may be asked to remain in the CRU until such abnormalities are deemed not clinically significant, or it is safe for outpatient follow-up.

A safety follow-up call will be made to participants approximately 28 to 35 days from administration of the final dose of study intervention.

# **Number of Participants**

Approximately 12 participants will be enrolled to study intervention.

Note: "Enrolled" means a participant's, or his or her legally authorized representative's, agreement to participate in a clinical study following completion of the informed consent process and screening. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol.

# **Intervention Groups and Duration**

Each participant will be screened to determine eligibility within 28 days prior to study treatment. Eligible participants will report to the CRU on Day -1 and will be required to stay in the CRU for 14 days and 13 nights. A safety follow-up call will be made to participants approximately 28 to 35 days from administration of the final dose of study intervention.

Each enrolled participant will participate in 2 study periods:

• Period 1: 300 mg PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses: Day 1 morning to Day 3 morning.

Period 2: 200 mg itraconazole, administered orally, QD, on Days 1 through 8, inclusive. On Days 4 through 6, participants will receive 300 mg
 PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses: Day 4 morning to Day 6 morning.

Participants will be discharged on Period 2, Day 9 following completion of all assessments.

The total planned duration of participation, from the Screening visit to the last Follow-up phone call, is approximately 10 weeks.

## Data Monitoring Committee or Other Independent Oversight Committee: No

#### **Statistical Methods**

# **Sample Size Determination**

A sample size of 9 participants will provide adequate precision to estimate the effects of itraconazole on the PK of PF-07321332. The expected widths of the 90% CIs with 80% coverage probability are shown in the following table for a range of possible effects.

| Parameter | <b>Estimated Effect</b> | 90% CI | CI Width |
|--------------------|-------------------------|------------|----------|
| | (100*Test/Reference) | | |
| AUC <sub>tau</sub> | 100% | 88%, 113% | 25% |
| | 110% | 97%, 124% | 27% |
| | 120% | 106%, 136% | 30% |
| | 130% | 115%, 147% | 32% |
| | 140% | 124%, 158% | 35% |
| $C_{max}$ | 100% | 92%, 108% | 16% |
| | 110% | 102%, 119% | 17% |
| | 120% | 111%, 130% | 19% |
| | 130% | 120%, 141% | 21% |
| | 140% | 129%, 152% | 22% |

These estimates are based on the assumption that within-participant standard deviations are 0.14 and 0.091 for  $lnAUC_{tau}$  and  $lnC_{max}$ , respectively, as obtained from ongoing clinical Study C4671001 in healthy participants.

To allow for dropouts, 12 participants will be enrolled in order to have 9 PK evaluable participants. Participants who withdraw from the study may be replaced at the discretion of the investigator upon consultation with the sponsor.

# **Pharmacokinetics Analysis**

The PK concentration population is defined as all participants who take at least 1 dose of study intervention and in whom at least 1 concentration value is reported.

The PK parameter analysis population is defined as all participants who take at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest are reported.

PK parameters for PF-07321332 will be analyzed using standard noncompartmental method of analysis. Actual PK sampling times will be used in the derivation of PF-07321332 PK parameters when available, otherwise nominal times will be used. The PF-07321332 PK parameters will be summarized descriptively by treatment and Day. Plasma concentrations will be listed and summarized descriptively by treatment, and nominal PK sampling time. Individual participant and summary profiles (mean and median plots) of the plasma concentration time data will be plotted using actual and nominal times, respectively. Box and whisker plots for AUC<sub>tau</sub> and C<sub>max</sub> following multiple doses of PF-07321332/ritonavir will be plotted by treatment.

## **Drug-Drug Interaction**

Natural log transformed AUC<sub>tau</sub>, and C<sub>max</sub> values of PF-07321332 will be analyzed using a mixed effect model with treatment as fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs will be obtained from the model. The adjusted mean differences and 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. PF-07321332/ritonavir administered alone will be the Reference treatment and PF-07321332/ritonavir co-administered with itraconazole will be the Test treatment.

#### **Safety Analysis**

AEs, ECGs, BP, RR, PR, and safety laboratory data will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of participants. Any clinical laboratory, ECG, BP, RR, and PR abnormalities of potential clinical concern will be described. Safety data will be presented in tabular and/or graphical format and summarized descriptively, where appropriate.

#### 1.2. Schema

| | Screening | Treatment | | |
|---|---|---|---|---|
| | | Period I | Period 2 | |
| | | Period I, Day -I to Day 4 | Period 2, Day 1 to Day 9 | |
| | | (Reference) PF-07321332/ritonavir 300 mg/100 mg q12h x 3 days (total of 5 doses) | (Test) Itraconazole:200 mg qd for 8 days + PF-07321332/ritonavir 300 mg/100 mg q12h x 3 days starting on Day 4 (total of 5 doses) | |
| Study<br>Days | Days -28 to -2 | Days -I to 4 | Days 5 to 13 | Days 28 to 35 |

#### 1.3. Schedule of Activities

The SoA table provides an overview of the protocol visits and procedures. Refer to the **STUDY ASSESSMENTS AND PROCEDURES** section of the protocol for detailed information on each procedure and assessment required for compliance with the protocol.

The investigator may schedule visits (unplanned visits) in addition to those listed in the SoA table, in order to conduct evaluations or assessments required to protect the well-being of the participant.

Period 1 (PF-07321332/ritonavir alone): Screening through Day 4

| Visit Identifier Abbreviations used in this table may be found in Appendix 8 | Screening <sup>a</sup> | Schedule for Period 1 | | | | |
|---|---|---|---|---|---|---|
| Days Relative to Day 1 | -28 to -2 | Day -1 | Day 1 | Day 2 | Day 3 | Day 4 |
| Informed consent | X | | | | | |
| CRU confinement <sup>b</sup> | | X | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ |
| Inclusion/exclusion criteria | X | X | | | | |
| Medical/medication history (update) <sup>c</sup> | X | X | | | | |
| Demography <sup>d</sup> | X | | | | | |
| Physical exame | X | X | | | | |
| Safety laboratory <sup>f</sup> | X | X | | | X | |
| CCI | | | | | | |
| FSHg | X | _ | | | _ | |
| Urine drug testing <sup>h</sup> | X | X | | | | |
| Serology: HBsAg, HBsAb, HBcAb, HCVAb, and HIV | X | | | | | |
| Pregnancy test (WOCBP only) | X | X | | | | |
| Contraception check <sup>i</sup> | X | X | | | | |
| 12-lead ECG (triplicate) <sup>j</sup> | X | | X | | X | |
| Vital signs (BP/PR/RR) <sup>k</sup> | X | | X | | X | |
| COVID-19 questionnaire <sup>1</sup> | X | X | | | | |
| COVID-19 testing <sup>m</sup> | X | X | | | | X |
| COVID-19 check temperature <sup>n</sup> | X | X | X | X | X | X |
| PF-07321332/ritonavir administration <sup>o</sup> | | · | X | X | X | |
| PK Blood Sampling for PF-07321332 and ritonavir <sup>p</sup> | | | X | X | X | X |
| Serious and non-serious AE monitoring | X | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ |

| Visit Identifier Abbreviations used in this table may be found in Appendix 8 | Screeninga | Schedule for Period 1 | | | | | |
|---|---|---|---|---|---|---|---|
| Prior and Concomitant Treatment(s) | X | $\rightarrow$ | _ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ |
| CCI | | | | | | | |

- a. Screening will be performed within 28 days prior to the first dose of PF-07321332/ritonavir.
- b. Participants will be admitted to the CRU on Day -1. Participants will be discharged on Day 13 following the final assessments.
- c. Medical history will include a history of prior illegal drug, alcohol, and tobacco use, as well as blood donation within prior 60 days. Medical history will be recorded at Screening and updated on Day -1 of Period 1.
- d. Demographics will include participant race, ethnicity, age, and gender during the Screening visit.
- e. A PE will be performed by trained medical personnel at the investigator site at Screening or Day -1 of Period 1 only (height and weight must be obtained at Screening to obtain BMI for eligibility criteria). A brief PE may be performed at other designated time points at the discretion of the investigator.
- f. Safety laboratory assessments including urinalysis, hematology, chemistry and coagulation will be performed at the indicated time-points. All the safety laboratory samples must be collected following at least a 4-hour fast. Additional safety laboratory assessments may be performed at any time at the discretion of the investigator.
- g. For postmenopausal (amenorrheic for at least 12 consecutive months) female participants only.
- h. Urine drug (mandatory) and alcohol breath test (at discretion of investigator) will be performed at Screening and on Day -1. These tests may be performed at any other time at the discretion of the investigator.
- i. The investigator or his/her designee will discuss with the participant the need to use highly effective contraception consistently and correctly according to contraception guidelines.
- j. Triplicate 12-lead ECG readings approximately 2 minutes apart will be taken at specified times. All ECG assessments will be made after at least a 5-minute rest in a supine position and prior to any blood draws or vital sign measurements.
- k. Single supine BP, RR and PR will be performed following at least a 5-minute rest in a supine position. BP, RR and PR assessments will be performed after collection of ECGs and prior to collection of blood draws if scheduled at the same time.
- 1. Check exposure to positive participant, residence or travel in area of high incidence and COVID-19 related signs and symptoms.
- m. The testing for COVID-19 pathogen by RT-PCR will be performed at each visit. For participants admitted for residence, a subsequent COVID-19 test will be performed after 4 days (ie, upon completion of 4 × 24 hours in house), or if they develop COVID-19 like symptoms.
- n. To be done at least daily during residence.
- o. PF-07321332/ritonavir will be administered orally, q12h for a total of 5 doses. PF-07321332 and ritonavir will be dosed simultaneously (within no more than 5 minutes of each other).
- p. One (approximately 4 mL) blood sample for PK analysis of PF-07321332 and ritonavir will be taken at the following timepoints: Day 1 predose the morning dose, Day 2 pre-dose the morning and evening doses, and Day 3 predose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, and 48 hours post the 5<sup>th</sup> dose of PF-07321332/ritonavir.

# Period 1 (PF-07321332/ritonavir alone): Detailed Sampling Schedule

| Visit Identifier | | Treatment Period | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | | | | | | | | | | | | 2 | | |
| Study Day | Da | y 1 | Da | y 2 | Day 3 | | | | | | | | Day<br>4 | Day<br>1 | | |
| Planned Hours Post Dose on that day | 0 | 12 | 0 | 12 | 0 | 0.5 | 1 | 1.5 | 2 | 4 | 6 | 8 | 12 | 16 | 24 | 48 |
| PF-07321332/ritonavir administration | X | X | X | X | X | | | | | | | | | | | |
| PK blood sampling | Xa | | Xa | Xa | Xa | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG (triplicate) | Xa | | | | Xa | | | X | | | | | | | | |
| Vital signs (BP/PR/RR) | Xa | | | | Xa | | | X | | | | | | | | |
| Safety laboratory | | | | | Xa | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | |

a. Predose sample collection.

# Period 2 (PF-07321332/ritonavir with itraconazole): Day 1 through Day 9

| Visit Identifier Abbreviations used in this table may be found in Appendix 8 | 1 | | Follow-Up | Early Termination/ Discontinuatio n | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Days Relative to Day 1 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | 28-35 Daysi | |
| CRU confinement | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | X | | | |
| Safety laboratory <sup>a</sup> | | | X | | | X | | | X | | X |
| CCI | | | | | | | | | | | |
| Contraception check | | | | | | | | | X | X | X |
| Pregnancy test (WOCBP only) | | | | | | | | | X | | X |
| 12-lead ECG (triplicate) <sup>b</sup> | X | | | X | | X | | | X | | X |
| Vital signs (BP/PR/RR) <sup>c</sup> | X | | | X | | X | | | X | | X |
| COVID-19 check temperature <sup>d</sup> | X | X | X | X | X | X | X | X | X | | |
| Itraconazole administration <sup>e</sup> | X | X | X | X | X | X | X | X | | | |
| PF-07321332/ritonavir administration <sup>f</sup> | | | | X | X | X | | | | | |
| PK Blood Sampling for PF-07321332 and ritonavir <sup>g</sup> | X | | | X | X | X | X | X | X | | X |
| Serious and non-serious adverse event monitoring | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | X | X |
| Concomitant treatment | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | X | X |
| Discharge from CRU <sup>h</sup> | | | | | | | | | X | | |

| Visit Identifier | | Schedule for Period 2 | | | | | | | | Follow-Up | Early |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Abbreviations used in this table may be found in | | | | | | | | | | | Termination/ |
| Appendix 8 | | | | | | | | | | | Discontinuatio |
| | | | | | | | | | | | n |
| Days Relative to Day 1 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | 28-35 Days <sup>i</sup> | |

- a. Safety laboratory assessments including urinalysis, hematology, chemistry, and coagulation. All the safety laboratory samples must be collected following at least a 4-hour fast. Additional safety laboratory assessments may be performed any time at the discretion of the Investigator.
- b. Triplicate 12-lead ECG readings approximately 2 minutes apart will be taken at specified times. All ECG assessments will be made after at least a 5-minute rest in a supine position and prior to any blood draws or vital sign measurements.
- c. Single supine blood pressure and pulse rate will be performed following at least a 5-minute rest in a supine position. BP and PR assessments will be performed after collection of ECGs and prior to collection of blood draws if planned together.
- d. To be done at least daily during residence.
- e. Participants will receive itraconazole 200 mg (in a 20 mL solution) once daily on Day 1 through Day 8.
- FF-07321332/ritonavir will be administered orally, q12h for a total of 5 doses. PF-07321332 and ritonavir will be dosed simultaneously (within no more than 5 minutes of each other).
- g. One (approximately 4 mL) blood sample for PK analysis of PF-07321332 will be taken at the following timepoints: Day 1 predose itraconazole dosing (48 hours post the last dose of PF-07321332 on Day 3), Day 4 predose the morning dose, Day 5 pre-dose the morning and evening doses, and Day 6 predose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, and 72 hours post the 5th dose of PF-07321332 celement.
- h. Participants will be eligible for discharge on Day 9 at the discretion of the investigator following PK sampling at 72 hours post the last dose of PF-07321332CCI
- i. Contact may occur via telephone and must occur 28 to 35 days from administration of the final dose of study intervention.

# Period 2 (PF-07321332/ritonavir with itraconazole): Detailed Sampling Schedule

| Visit Identifier | | Treatment Period | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period 2 Study Day | Day<br>1 | Da | ıy 4 | Da | Day 5 Day 6 Day Day 1 7 8 | | | | | | | | Day<br>9 | | | | | |
| Planned Hours Post Dose on that day | 0 | 0 | 12 | 0 | 12 | 0 | 0.5 | 1 | 1.5 | 2 | 4 | 6 | 8 | 12 | 16 | 24 | 48 | 72 |
| PF-07321332/ritonavir administration | | X | X | X | X | X | | | | | | | | | | | | |
| Itraconazole administration | X | X | | X | | X | | | | | | | | | | X | X | |
| PK blood sampling | Xa | Xa | | Xa | Xa | Xa | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG (triplicate) | Xa | Xa | | | | Xa | | X | X | | | | | | | | | X |
| Vital signs (BP/PR/RR) | Xa | Xa | | | | Xa | | X | X | | | | | | | | | X |
| CCI | | | | | | | | | | | | | | | | | | |
| Safety laboratory | | | | | | Xa | | | | | | | | | | | | X |

a. Predose itraconazole administration on Day 1; predose PF-07321332/ritonavir administration on Days 4, 5, and 6.

#### 2. INTRODUCTION

PF-07321332 is a potent and selective inhibitor of the SARS-CoV-2 3CL protease that is currently being developed as an oral treatment of COVID-19. Ritonavir is a strong CYP3A4 inhibitor being used to inhibit the metabolism of PF-07321332 in order to increase plasma concentrations of PF-07321332 to values that are anticipated to be efficacious.

## 2.1. Study Rationale

The purpose of the study is to evaluate the effect of the strong CYP3A4 inhibitor, itraconazole, on the PK of PF-07321332 in healthy participants. Results from this study will provide guidance for dosing recommendations with concomitant medications during Phase 3 development and further establish the safety margins of PF-07321332/ritonavir.

# 2.2. Background

In December 2019, COVID-19 was identified as a new, potentially fatal, respiratory infection caused by the novel coronavirus, SARS-CoV-2. The WHO declared COVID-19 a Public Health Emergency of International Concern on 20 January 2020 and further characterized the disease outbreak as a pandemic on 11 March 2020.<sup>2</sup>

PF-07321332 is an orally bioavailable  $3CL^{pro}$  inhibitor shown to be effective against SARS-CoV-2  $3CL^{pro}$  ( $K_i$  = 0.00311  $\mu$ M) in a biochemical enzymatic assay. Since the  $3CL^{pro}$  from human coronaviruses are structurally similar and share a high degree of conservation at the active site of the enzyme, the ability of PF-07321332 to inhibit the  $3CL^{pro}$  of other coronaviruses (SARS-CoV-1 and HCoV-229E, MERS, HCoV-OC43, HCoV-HKU1, and HCoV-NL63) was also confirmed, indicating a potential for broad spectrum anti-coronavirus activity. The coronavirus 3CL protease is a virally encoded enzyme that is critical to the SARS-CoV-2 replication cycle, analogous to other obligatory virally encoded proteases (eg, HIV Protease, HCV Protease). PF-07321332 is being developed as an oral treatment in patients with COVID-19 infection.

Ritonavir is a strong CYP3A4 inhibitor being used to inhibit the metabolism of PF-07321332 in order to increase plasma concentrations of PF-07321332 to values that are anticipated to be efficacious. Ritonavir is not expected to have any pharmacological impact on the SARS-CoV-2 virus and its elimination is not expected to be significantly altered by renal impairment. Ritonavir is being used only as a PK boosting agent.

#### 2.2.1. Nonclinical Pharmacology

Details of the nonclinical pharmacology of PF-07321332 can be found in the current IB.

# 2.2.2. Nonclinical Pharmacokinetics and Metabolism

Hepatic CYP3450 enzymes were identified as the main pathway for clearance of PF-07321332 in vitro in liver microsomes (mouse, rat, hamster, rabbit, monkey, and human), hepatocytes (rat, monkey, and human), and in vivo in rat and monkey after repeat oral dosing. In a reaction phenotyping study using human liver microsomes in the presence of

PFIZER CONFIDENTIAL

selective CYP inhibitors, CYP3A4 was predicted to be the major contributor ( $f_m = 0.99$ ) to the in vitro oxidative metabolism of PF-07321332. No significant CYP3A5 contribution is expected to the metabolism of PF-07321332. Urinary excretion of PF-07321332 following single IV or oral doses in rats was approximately 11%, suggesting minor urinary contributions to the overall elimination of PF-07321332.

Additional information of the nonclinical PK and metabolism of PF-07321332 is available in the current IB.

## 2.2.3. Nonclinical Safety

There were no adverse findings observed in repeat-dose toxicity studies in rats and monkeys up to two weeks duration and the NOAELs were the highest dose administered (1000 mg/kg and 600 mg/kg in the rat and monkey studies, respectively). PF-07321332-related non-adverse, test article-related clinical findings included sporadic occurrence of emesis with slight body weight decreases in monkeys. Monitorable and reversible clinical pathology findings included those possibly suggestive of low-grade inflammation (in rats and monkeys) or alterations in the coagulation pathways (in rats only) without clinical or microscopic correlates. Other non-adverse clinical pathology findings were likely due to the emesis and subsequent dehydration in monkeys. In rats administered 1000 mg/kg/day, lower mean absolute and relative heart weights (females) and higher absolute and relative liver weights (both sexes) were observed relative to controls. The lower heart weights had no microscopic correlates and were fully reversed at the end of the 2-week recovery period. Higher liver weights correlated with reversible, non-adverse microscopic findings of minimal to mild severity in the liver and thyroid gland consistent with adaptive changes related to microsomal enzyme induction.

PF-07321332 was not mutagenic or clastogenic in in vitro genetic toxicity studies and was negative in the in vivo rat micronucleus assay incorporated into the GLP repeat-dose rat toxicity study.

The nonclinical studies performed adequately support the oral administration of PF-07321332 in the clinic for up to 14 days.

Further details of the nonclinical safety program are provided in the current IB.

#### 2.2.4. Clinical Overview

Safety, tolerability and PK of PF-07321332 in healthy adult participants is currently being explored in an ongoing Phase 1 FIH Study (C4671001). Study C4671001 is a four-part study consisting of SAD (PART-1), MAD (PART-2), relative bioavailability/food effect (PART-3), and metabolism and excretion study (PART-4). PART-1 and -2 are randomized, double-blind, sponsor-open, and placebo-controlled to evaluate safety, tolerability, and PK of single and multiple escalating oral doses of PF-07321332, respectively. PART-3 is randomized and open-label to evaluate relative bioavailability and food effect of an oral tablet formulation. PART-4 is open-label, non-randomized, single-period to evaluate the

metabolism and excretion of PF-07321332. Included in this Clinical Overview are summaries of the preliminary results from PART-1 and PART-2.

# 2.2.4.1. Safety Overview

Preliminary safety and tolerability data from Study C4671001 as of 7 April 2021 in PART-1 and 14 April 2021 in PART-2 (data snapshot taken) demonstrated PF-07321332 was generally safe and well-tolerated in healthy participants at single doses of PF-07321332 ranging from 150 mg to 1500 mg alone and at 250 mg and 750 mg with ritonavir (100 mg at -12h, 0h, 12h) in the PART-1: SAD, and ten days of dosing from 75 mg q12h to 500 mg q12h with 100 mg ritonavir q12h in the PART-2: MAD of the study.

Following single doses of PF-07321332 with and without ritonavir, all AEs were mild and none were considered treatment related. There were no obvious trends in, or association of, TEAEs with dose level of PF-07321332. Following multiple doses, the most commonly observed AEs by system organ class were gastrointestinal disorders and nervous system disorders. Diarrhea was the most common reported AE, occurring in 4 participants across treatment groups. A total of 5 treatment related TEAEs were observed in Part-2:MAD. Across treatment groups, blood TSH increased in 3 participants, and 2 participants reported dysgeusia. The 3 participants with elevated TSH results did not experience related clinical symptoms and the free T4 results remained within reference range.

Based on review of preliminary (unaudited) data, all reported adverse events have been of mild intensity. There have been no deaths, serious adverse events, or SUSARs reported. There were no clinically meaningful findings in vital signs, ECG, or potential Hy's Law cases reported during this study.

Further details on the clinical safety information with PF-07321332 are provided in the current IB.





#### 2.3. Benefit/Risk Assessment

PF-07321332/ritonavir or itraconazole are not expected to provide any clinical benefit to healthy participants in this study. This study is designed primarily to estimate the effect of multiple doses of itraconazole on the PK of PF-07321332 to provide guidance for dosing recommendations with concomitant medications for PF-07321332/ritonavir.



More detailed information about the known and expected benefits and risks and reasonably expected adverse events of PF-07321332 may be found in the IB, which is the SRSD for PF-07321332. The SRSDs for ritonavir<sup>4</sup> and itraconazole<sup>5</sup> are the corresponding SmPCs.

# 2.3.1. Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | Study Intervention(s): PF-07321332 | |
| Emesis | Sporadic emesis was observed at ≥100 mg/kg/day of PF-07321332 in the 15-day NHP toxicology study (See IB). Based on preliminary data, no emesis was observed in the FIH Study C4671001 at single doses of PF-07321332 up to 1500 mg alone and up to 750 mg administered with ritonavir (100 mg at -12h, 0h, 12h), and at repeated daily doses administered orally for ten days of up to 500 mg PF-07321332 q12h with 100 mg ritonavir q12h. | As this is an investigational agent, there is some risk that is mitigated by close observation of AEs, etc. If needed, palliative care or antiemetics may be provided. |
| Neuronal and pulmonary effects | Transient effect in rat neuronal and pulmonary endpoints were observed in rat toxicology study at the high dose level (1000 mg/kg as single dose; See IB). Based on preliminary data, no AEs suggestive of neuronal or pulmonary effects were observed in the FIH Study C4671001 at single doses of PF-07321332 up to 1500 mg alone and up to 750 mg administered with ritonavir (100 mg at -12h, 0h, 12h), and at repeated daily doses administered orally for ten days of up to 500 mg PF-07321332 q12h with 100 mg ritonavir q12h. | Vital signs, including respiratory rate, will be monitored for pulmonary effect. There will be close observation of AEs for any signs of neuronal effect. |
| Hemodynamic effects | Low level inflammation (increase in fibrinogen) in 15-day NHP toxicology study and changes in platelets, globulin and albumin/globulin ratio and coagulation system (increase in PT and aPTT) in 14-day rat toxicology study (See IB). No relevant laboratory changes in inflammatory markers have been observed in the FIH Study C4671001 at single doses of PF-07321332 up to 1500 mg alone and up to 750 mg administered with ritonavir (100 mg at -12h, 0h, 12h), and at repeated daily doses administered orally for ten days of up to 500 mg PF-07321332 q12h with 100 mg ritonavir q12h. | Fibrinogen, platelets, PT-INR and aPTT, albumin and total proteins will be monitored. |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Thyroid function studies | In 14-day rat toxicology study at high dose of PF-07321332 (1000 mg/kg/day) thyroid gland changes observed were of low severity and without evidence of tissue damage. In the FIH Study C4671001, 3 participants had TEAEs of elevated TSH levels across treatment groups (PF-07321332 or placebo with ritonavir 100 mg q12h) in the MAD part of the study. There was no clinical correlation with these TSH changes and free T4 remained within reference range at all times. | TSH and free T4 will be evaluated to monitor thyroid function |
| | Study Intervention(s): Ritonavir | |
| Gastrointestinal disturbances (including diarrhea, nausea, vomiting and abdominal pain). | Frequently reported adverse reaction in HIV patients at 600 mg BID. | Lower dose of 100 mg twice daily is used in this study. There will be close observation of AEs. If needed, anti-emetics may be provided. |
| Neurological disturbances (eg, paresthesia, including oral paresthesia, dysgeusia and dizziness). | Frequently reported adverse reaction in HIV patients at 600 mg BID. | Lower dose used in this study. There will be close observation of AEs. |
| Rash (most commonly reported as erythematous and maculopapular, followed by pruritic). | Frequently reported adverse reaction in HIV patients at 600 mg BID. | Lower dose used in this study. There will be close observation of AEs and monitoring through targeted physical exams. If needed, palliative care may be provided. |
| Fatigue/Asthenia. | Frequently reported adverse reaction in HIV patients at 600 mg BID. | Lower dose used in this study. There will be close observation of AEs and monitoring through targeted physical exams. |
| Limited case reports of renal toxicity | Although ritonavir therapy is not generally considered nephrotoxic, a limited number of cases of acute kidney injury secondary to ritonavir have been reported postmarketing in HIV patients. | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Intervention(s) Itraconazole | | |
| Hepatotoxicity | Itraconazole has been associated with rare cases of serious hepatotoxicity, including liver failure and death. Some of these cases had neither pre-existing liver disease nor a serious underlying medical condition, and some of these cases developed within the first week of treatment. If clinical signs or symptoms develop that are consistent with liver disease, treatment should be discontinued, and liver function testing performed. | Short-term or intermittent dosing with itraconazole (eg less than 14 days), is generally considered to be associated with a lower risk of liver injury relative to chronic dosing. Liver function will be monitored. |
| Cardiac dysrhythmias | Life-threatening cardiac dysrhythmias and/or sudden death have occurred in patients using drugs such as cisapride, pimozide, methadone, or quinidine concomitantly with itraconazole and/or other CYP3A4 inhibitors. | Short-term dosing of itraconazole will be used in this study. Concomitant use of prescription and non-prescription drugs are not allowed. Participants with underlying cardiac disease will be excluded. Cardiac function will be monitored. |
| Reports of congestive heart failure | Itraconazole has been associated with reports of congestive heart failure. In post-marketing experience, heart failure was more frequently reported in patients receiving a total daily dose of 400 mg although there were also cases reported among those receiving lower total daily doses. | This study will utilize a dose of 200 mg daily. Participants with risk factors for congestive heart failure are excluded. Cardiac function will be monitored. |

#### 2.3.2. Benefit Assessment

PF-07321332/ritonavir and itraconazole will not provide any clinical benefit to healthy participants in this study. Any anticipated benefit to participants would be in terms of contribution to the process of developing a new therapy in an area of unmet medical need.

#### 2.3.3. Overall Benefit/Risk Conclusion

PF-07321332/ritonavir and itraconazole are not expected to provide any clinical benefit to healthy participants in this study. Taking into account the measures taken to minimize risk to participants of this study, the potential risks identified in association with administration of PF-07321332/ritonavir and itraconazole are justified by the anticipated benefit, in terms of contribution to the process of developing a new therapy in an area of unmet medical need.

## 3. OBJECTIVES AND ENDPOINTS

| Primary Objective: | Primary Endpoint: |
|---|---|
| To estimate the effect of multiple doses of itraconazole on the PK of PF-07321332 following multiple doses of PF-07321332/ritonavir | PF-07321332 plasma PK parameters: C <sub>max</sub> and AUC <sub>tau</sub> with itraconazole (test) versus without itraconazole (reference) |
| Secondary Objective: | Secondary Endpoints: |
| <ul> <li>To evaluate the safety and tolerability of PF-07321332/ritonavir in healthy participants in the absence and presence of multiple doses of itraconazole</li> <li>To characterize the PK of PF-07321332 following multiple doses when PF-07321332/ritonavir is administered alone or with itraconazole in healthy participants.</li> </ul> | <ul> <li>Assessment of TEAEs, clinical laboratory abnormalities, vital signs, physical exam, and 12-lead ECGs</li> <li>PF-07321332 plasma PK parameters: T<sub>max</sub>, t<sub>1/2</sub>, AUC<sub>last</sub>, CL/F, and V<sub>z</sub>/F for PF-07321332 with and without coadministration of itraconazole.</li> </ul> |

#### 4. STUDY DESIGN

# 4.1. Overall Design

This is a Phase 1, open-label, 2-period, fixed-sequence crossover study to estimate the effect of the strong CYP3A4 inhibitor, itraconazole, on the PK of PF-07321332 in healthy participants. The study will consist of 2 treatments: multiple oral doses of 300 mg PF-07321332/100 mg ritonavir alone and multiple oral doses of 300 mg PF-07321332/100 mg ritonavir in combination with itraconazole. A total of approximately 12 healthy male and/or female participants will be enrolled into the study to ensure at least 9 participants will complete the study. The treatment will consist of a single-fixed sequence.

Participants who discontinue from the study for non-safety reasons may be replaced at the sponsor's discretion in collaboration with the Investigator.

Healthy participants will be screened to determine eligibility within 28 days prior to study treatment. Medical history and results of physical examination, physical measurements, vital signs, 12-lead ECGs, and clinical laboratory evaluations will determine eligibility. Participants will report to the CRU on Day -1, at least 12 hours prior to Day 1 dosing in Period 1 and will be required to stay in the CRU for 14 days and 13 nights.

In Period 1, each enrolled participant will receive 300 mg PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses, from Day 1 morning to Day 3 morning. Serial PK samples will be collected up to 48 hours post the 5<sup>th</sup> dose on Day 3 to establish baseline exposure of PF-07321332 and ritonavir. PK samples will also be collected predose the morning and evening doses of PF-07321332/ritonavir on Day 2 to confirm steady state.

Period 2 will begin on Study Day 5 (referred to as Period 2, Day 1). Participants will receive 200 mg itraconazole, administered orally, QD on Period 2, Days 1 through 8, inclusive. On Days 4, 5, and 6, participants will receive 300 mg PF-07321332/100 mg ritonavir administered orally, q12h for 5 doses, from Day 4 morning to Day 6 morning. Following the final administration of PF-07321332/ritonavir on the morning of Day 6, participants will undergo serial PK sampling up to 72 hours post the last dose. PK samples will also be collected predose the morning and evening doses of PF-07321332/ritonavir on Day 5 to confirm steady state. Participants will be discharged from the CRU on Day 9 (Study Day 13) following completion of all assessments.

If a participant has any clinically significant, study related abnormalities at the conclusion of a scheduled inpatient portion of the study, the Pfizer medical monitor (or designated representative) should be notified and the participant may be asked to remain in the CRU until such abnormalities are deemed not clinically significant, or it is safe for outpatient follow-up.

A safety follow-up call will be made to participants approximately 28 to 35 days from administration of the final dose of study intervention.

The total planned duration of participation, from the Screening visit to the last Follow-up phone call, is approximately 10 weeks.

# 4.2. Scientific Rationale for Study Design

In vitro and in vivo metabolite profiling suggests that the primary clearance mechanism for PF-07321332 is CYP3A4 mediated oxidation ( $f_m = 0.99$ ). As such, in the FIH Study, C4671001, the CYP3A4 inhibitor ritonavir was used to enhance the exposure of PF-07321332 in order to achieve plasma levels that are anticipated to be efficacious. Preliminary PK data following multiple oral administrations of PF-07321332/ritonavir at doses ranging from 75/100 mg to 500/100 mg q12h suggest that the renal pathway may also play a significant role in PF-07321332 excretion when co-administered with ritonavir (32.5%)

to 64.6% of the drug excreted unchanged in urine across doses at steady-state). Ritonavir is extensively metabolized, primarily by CYP3A4. Mechanistically, inhibition of CYP3A4 could further decrease the metabolism of PF-07321332 and ritonavir, and thereby increase circulating exposures. The objective of this study is to evaluate the effect of a probe CYP3A4 inhibitor, at steady-state, on the pharmacokinetics, safety and tolerability of PF-07321332/ritonavir.

The inhibitor to be utilized in this study is itraconazole. Itraconazole and its primary metabolite (hydroxy-itraconazole) are specific strong inhibitors of CYP3A. For these characteristics, along with its safety profile, itraconazole has often been utilized as a perpetrator drug for CYP3A inhibition PK drug interaction studies. Since PF-07321332 and ritonavir are substrates of CYP3A, concomitant administration of multiple doses (to reach steady state levels) of itraconazole along with PF-07321332/ritonavir may lead to increased systemic exposure of PF-07321332 and ritonavir. This may require PF-07321332/ritonavir dose adjustment when it is utilized with medications that are strong CYP3A inhibitors. Results of this study will provide guidance for dosing recommendations with concomitant medications and further establish the safety margins of PF-07321332/ritonavir.

## 4.2.1. Choice of Contraception/Barrier Requirements

Human reproductive safety data are limited for PF-07321332, but there is no suspicion of human teratogenicity based on the intended pharmacology of the compound. Therefore, the use of a highly effective method of contraception is required (see Appendix 4).

## 4.2.2. Collection of Retained Research Samples

Retained Research Samples will be collected and stored for further analyses which may, for example, provide greater understanding of the study intervention.

## 4.3. Justification for Dose

This study is designed to estimate the effect of multiple dose administration of 200 mg daily itraconazole on multiple dose PK of PF-07321332 and ritonavir. A dose of 300 mg PF-07321332, pharmacokinetically enhanced with 100 mg ritonavir, to be administered q12h for 5 doses with and without itraconazole will be used. This dose is the intended therapeutic dose to be evaluated in Phase 2/3 studies and is appropriate considering concomitant administration of PF-07321332 with ritonavir provides near maximal CYP3A4 inhibition and the addition of itraconazole is not expected to result in a significant increase of systemic exposures of PF-07321332.

An oral dose of itraconazole 200 mg solution administered QD for 8 days will be used to provide a substantial degree of CYP3A4 inhibition. Doses greater than 200 mg are not

expected to provide any additional CYP3A4 inhibition. PF-07321332/ritonavir will be administered under fasting conditions approximately 1 hour after itraconazole administration on Period 2, Days 4, 5, and 6 to maximize itraconazole systemic exposures and CYP3A4 inhibition. Itraconazole will continue to be administered on Period 2, Days 7 and 8 to maintain maximal CYP3A4 inhibition until completion of PK sampling.

# 4.4. End of Study Definition

The end of the study is defined as the date of last scheduled procedure shown in the SoA for the last participant in the trial.

A participant is considered to have completed the study if he/she has completed all parts of the study, including the last scheduled procedure shown in the SoA.

#### 5. STUDY POPULATION

This study can fulfill its objectives only if appropriate participants are enrolled. The following eligibility criteria are designed to select participants for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular participant is suitable for this protocol.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

# Age and Sex:

- 1. Participants must be 18 to 60 years of age, inclusive, at the time of signing the ICD.
  - Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

# **Type of Participant and Disease Characteristics:**

- 2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, PE, laboratory tests, vital signs and standard 12-lead ECGs.
- 3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
- 4. Female participants must have a negative pregnancy test.

# Weight:

5. BMI of 17.5 to  $30.5 \text{ kg/m}^2$ ; and a total body weight >50 kg (110 lb).

#### **Informed Consent:**

6. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

#### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions:**

- 1. Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
- 2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
- 3. Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy- or brady-arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than NYHA 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
- 4. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
- 5. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
- 6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

# **Prior/Concomitant Therapy:**

7. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention. Refer to Section 6.8 Concomitant Therapy for additional details.

- 8. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s). Refer to Section 6.8 Concomitant Therapy.
- 9. Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.

# **Prior/Concurrent Clinical Study Experience:**

10. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

# **Diagnostic Assessments:**

- 11. A positive urine drug test.
- 12. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
- 13. Baseline 12-lead ECG (triplicate) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant. The average of triplicate measurement should be used for eligibility determination.
- 14. Participants with <u>ANY</u> of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:
  - AST or ALT level  $> 1.0 \times ULN$ ;
  - Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

• eGFR < 81 mL/min/1.73 m<sup>2</sup> (eg <90 mL/min/1.73 m<sup>2</sup> with 10% variation) based on the CKD-EPI equation.

#### **Other Exclusions:**

- 15. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
- 16. Use of tobacco or nicotine containing products in excess of the equivalents of 5 cigarettes per day or 2 chews of tobacco per day.
- 17. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
- 18. History of sensitivity to heparin or heparin-induced thrombocytopenia.
- 19. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
- 20. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
- 21. History of sensitivity reactions to ritonavir or itraconazole, or any of the formulation components of PF-07321332, ritonavir, or itraconazole.
- 22. Pregnant or breastfeeding women.

#### 5.3. Lifestyle Considerations

The following guidelines are provided:

#### 5.3.1. Meals and Dietary Restrictions

- Participants must abstain from all food and drink (except water) at least 4 hours prior to any safety laboratory evaluations and 10 hours prior to drug administration for:
  - o Dosing of itraconazole on Period 2, Day 4, Day 5, and Day 6
  - Morning PF-07321332/ritonavir administration on Period 1, Day 3 and Period 2, Day 6.
- At least a 2-hour fast is required prior to drug administration for:
  - o Evening dosing of PF-07321332/ritonavir in Periods 1 and 2

- o Morning dosing of PF-07321332/ritonavir on Period 1, Days 1 and 2
- o Itraconazole dosing on Period 2, Day 1 to Day 3, and Days 7 and 8.
- A light breakfast is permitted 2 hours after dosing on non-PK days. On PK days (Period 1, Day 3 and Period 2, Day 6), no food will be permitted for 4 hours after dosing.
- Water is permitted until 1 hour prior to study intervention administration. Water
  consumption is not restricted after evening doses on PK days and after all doses on
  non-PK days. Water may be consumed without restriction beginning 1 hour after
  PF-07321332/ritonavir morning dosing on PK days. Noncaffeinated drinks (except
  grapefruit or grapefruit-related citrus fruit juices—see below) may be consumed with
  meals and the evening snack.
- Lunch will be provided approximately 4 hours after the last dose of the morning of either itraconazole or PF-07321332/ritonavir.
- Dinner will be provided approximately 9 to 10 hours after the last dose of the morning of either itraconazole or PF-07321332/ritonavir.
- An evening snack may be permitted.
- Participants will refrain from consuming red wine, grapefruit, or grapefruit-related citrus fruits (eg, Seville oranges, pomelos, fruit juices) from 7 days prior to the first dose of study intervention until collection of the final PK blood sample.
- While participants are confined, their total daily nutritional composition should be approximately 55% carbohydrate, 30% fat, and 15% protein. The daily caloric intake per participant should not exceed approximately 3200 kcal.

#### 5.3.2. Caffeine, Alcohol, and Tobacco

- Participants will abstain from caffeine-containing products for 24 hours prior to the start of dosing until collection of the final PK sample of each study period.
- Participants will abstain from alcohol for 24 hours prior to admission (except as stated above for red wine) to the CRU and continue abstaining from alcohol until collection of the final PK sample of each study period. Participants may undergo an alcohol breath test or blood alcohol test at the discretion of the investigator.
- Participants will abstain from the use of tobacco- or nicotine-containing products for 24 hours prior to dosing and during confinement in the CRU.

# **5.3.3.** Activity

- Participants will abstain from strenuous exercise (eg, heavy lifting, weight training, calisthenics, aerobics) for at least 48 hours prior to each blood collection for clinical laboratory tests. Walking at a normal pace will be permitted;
- In order to standardize the conditions on PK sampling days, participants will be required to refrain from lying down (except when required for BP, PR, RR, and ECG measurements) for first 4 hours after morning dose, and may be required to follow meals and dietary restrictions.

# **5.3.4.** Contraception

The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant and his or her partner(s) from the permitted list of contraception methods (see Appendix 4 Section 10.4.4) and will confirm that the participant has been instructed in its consistent and correct use. At time points indicated in the schedule of activities (SoA), the investigator or designee will inform the participant of the need to use highly effective contraception consistently and correctly and document the conversation and the participant's affirmation in the participant's chart (participants need to affirm their consistent and correct use of at least 1 of the selected methods of contraception) considering that their risk for pregnancy may have changed since the last visit. In addition, the investigator or designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant or partner.

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently enrolled in the study. Screen failure data are collected and remain as source and are not reported on the CRF.

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened.

# 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, medical device(s), or study procedure(s) intended to be administered to a study participant according to the study protocol.

For the purposes of this protocol, study intervention refers to PF-07321332, ritonavir and itraconazole.

# 6.1. Study Intervention(s) Administered

PF-07321332 will be provided by Pfizer as bulk powders for extemporaneous preparation of oral suspensions at the CRU.

PF-07321332 will be presented to the participants in individual dosing containers.

Ritonavir (Norvir® or other local commercialized product) 100 mg tablets will be supplied locally by the CRU.

Itraconazole (Sporanox®) oral solution 10 mg/mL will be supplied by the CRU.

#### **6.1.1.** Administration

Investigational products will be administered orally and according to the conditions described in the SoA section and Protocol Section 5.3.1 Meals and Dietary Restrictions.

In Period 1, Day 1 following an overnight fast of at least 10 hours, participants will receive 300 mg PF-07321332, administered orally with 100 mg ritonavir (as 1 × 100 mg tablet) administered orally starting at approximately 0800 hours (plus or minus 2 hours). PF-07321332 and ritonavir will be dosed simultaneously (within no more than 5 minutes of each other). Participants will receive 300 mg PF-07321332, with 100 mg ritonavir (as 1 × 100 mg tablet) administered orally every 12 hours for a total of 5 doses, with the last dose administered on the morning of Day 3. On Day 3, PF-07321332/ritonavir dose should be administered following an overnight fast of at least 10 hours. At least a 2-hour fast is required for evening dosing. Participants will swallow ritonavir tablets whole and will not chew prior to swallowing.

Investigator site personnel will administer study intervention with ambient temperature water to a total volume of approximately 240 mL. Study intervention will be administered according to the EDR and the protocol.

In Period 2, Days 1 through 8, participants will receive itraconazole oral solution dose of 200 mg at approximately 0800 hours (plus or minus 2 hours). Investigator site personnel will administer itraconazole with ambient temperature water to a total volume of approximately 240 mL. Approximately 1 hour after the itraconazole dose on Days 4 through 6, participants will receive 300 mg PF-07321332 with 100 mg ritonavir (as 1 × 100 mg tablet), both administered orally, starting at approximately 0900 hours (plus or minus 2 hours). Participants will receive 300 mg PF-07321332, with 100 mg ritonavir (as 1 × 100 mg tablet) administered orally every 12 hours on Days 4 through 6, for a total of 5 doses, starting with the first dose on the morning of Period 2, Day 4 and the last dose administered on the morning of Day 6. On Days 4 through 6, itraconazole should be administered following an overnight fast of at least 10 hours. At least a 2-hour fast is required for evening dosing of PF-07321332/ritonavir and for itraconazole dosing on all other days. PF-07321332 and ritonavir will be dosed simultaneously (within no more than 5 minutes of each other).

Commercial itraconazole (Sporanox®) oral solution will be dispensed at the CRU into oral syringes by 2 operators, one of whom is an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, practitioner, or pharmacist) as

allowed by local, state, and institutional guidance. Investigator site personnel will administer study intervention with ambient temperature water to a total volume of approximately 240 mL. Study intervention will be administered according to the EDR and the protocol.

| Intervention Name | PF-07321332 | Ritonavir | Itraconazole |
|---|---|---|---|
| Туре | Drug | Boosting agent | CYP3A4 index inhibitor |
| Dose Formulation | Suspension | Tablet | Solution |
| Unit Dose Strength(s) | N/A | 100 mg | 10 mg/mL |
| Dosage Level(s) | 300 mg | 100 mg | 200 mg |
| Route of<br>Administration | Oral | Oral | Oral |
| Use | Experimental | PK Boosting agent | CYP3A4 index inhibitor |
| IMP or NIMP | IMP | NIMP | NIMP |

# 6.2. Preparation, Handling, Storage, and Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study interventions received and any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study interventions must be stored in a secure, environmentally controlled, and monitored (manual or automated recording) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff. At a minimum, daily minimum and maximum temperatures for all site storage locations must be documented and available upon request. Data for nonworking days must indicate the minimum and maximum temperatures since previously documented for all site storage locations upon return to business.
- 3. Any excursions from the study intervention label storage conditions should be reported to Pfizer upon discovery along with any actions taken. The site should actively pursue options for returning the study intervention to the storage conditions described in the labeling, as soon as possible. Once an excursion is identified, the study intervention must be quarantined and not used until Pfizer provides permission to use the study intervention. Specific details regarding the definition of an excursion and information the site should report for each excursion will be provided to the site in the PCRU site procedures.
- 4. Any storage conditions stated in the SRSD will be superseded by the storage conditions stated on the label.
- 5. Study interventions should be stored in their original containers.

- 6. See the EDR for storage conditions of the PF-07321332. See the ritonavir and itraconazole package insert for storage conditions of the study intervention prior to and after preparation.
- 7. The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records), such as the IPAL or sponsor-approved equivalent. All study interventions will be accounted for using a study intervention accountability form/record.
- 8. Further guidance and information for the final disposition of unused study interventions are provided in the PCRU's site procedures. All destruction must be adequately documented. If destruction is authorized to take place at the investigator site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer.

Upon identification of a product complaint, notify the sponsor within 1 business day of discovery.

# 6.2.1. Preparation and Dispensing

Within this protocol, preparation refers to the investigator site activities performed to make the study intervention ready for administration or dispensing to the participant by qualified staff. Dispensing is defined as the provision of study intervention, concomitant treatments, and accompanying information by qualified staff member(s) to a healthcare provider, participant in accordance with this protocol. Local health authority regulations or investigator site guidelines may use alternative terms for these activities.

See the EDR for PF-07321332 for instructions on how to prepare the study intervention for administration. Commercial ritonavir (Norvir® or other local commercialized product) oral tablet will be dispensed at the CRU into individual dosing containers using the package insert as guidance. Commercial itraconazole (Sporanox®) oral solution will be dispensed at the CRU into oral syringes using the package insert as guidance. All study intervention should be prepared and dispensed by an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacy assistant/technician, or pharmacist) as allowed by local, state, and institutional guidance. A second staff member will verify the dispensing.

# 6.3. Measures to Minimize Bias: Randomization and Blinding

# 6.3.1. Allocation to Study Intervention

The investigator will assign participant numbers to the participants as they are screened for the study.
## 6.4. Study Intervention Compliance

When participants are dosed at the site, they will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of each dose administered in the CRU will be recorded in the source documents and recorded in the CRF. The dose of study intervention and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention. Study site personnel will examine each participant's mouth to ensure that the study intervention was ingested.

#### 6.5. Dose Modification

No dose modification is anticipated.

## 6.6. Continued Access to Study Intervention After the End of the Study

No intervention will be provided to study participants at the end of their study participation.

#### 6.7. Treatment of Overdose

For this study, any dose of PF-07321332 greater than 600 mg, ritonavir 200 mg, or itraconazole 200 mg within a 24-hour time period [±2 hours] will be considered an overdose.

There is no specific treatment for an overdose.

In the event of an overdose, the investigator should:

- 1. Contact the medical monitor within 24 hours.
- 2. Closely monitor the participant for any AEs/SAEs and laboratory abnormalities for at least 5 half-lives or 28 calendar days after the overdose of PF-07321332/ritonavir or itraconazole (whichever is longer).
- 3. Document the quantity of the excess dose as well as the duration of the overdose in the CRF.
- 4. Overdose is reportable to Pfizer Safety only when associated with an SAE.
- 5. Obtain a blood sample for PK analysis within 1 day from the date of the last dose of study intervention if requested by the medical monitor (determined on a case-by-case basis).

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the medical monitor based on the clinical evaluation of the participant.

## 6.8. Concomitant Therapy

Use of prescription or nonprescription drugs and dietary and herbal supplements are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study

intervention. Limited use of nonprescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor. Acetaminophen/paracetamol may be used at doses of  $\leq 1$  g/day.

Hormonal contraceptives that meet the requirements of this study are allowed to be used in participants who are WOCBP (see Appendix 4).

All concomitant treatments taken during the study must be recorded with indication, daily dose, and start and stop dates of administration. All participants will be questioned about concomitant treatment at each site visit.

Treatments taken within 28 days before the first dose of study intervention will be documented as a prior treatment. Treatments taken after the first dose of study intervention will be documented as concomitant treatments.

#### 6.8.1. Rescue Medicine

There is no rescue therapy to reverse the AEs observed with PF-07321332, ritonavir, or itraconazole; standard medical supportive care must be provided to manage the AEs.

# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Intervention

It may be necessary for a participant to permanently discontinue study intervention. Reasons for permanent discontinuation of study intervention include the following.

- AE requiring discontinuation in investigator's view;
- Pregnancy;
- Positive COVID-19 test.

If study intervention is permanently discontinued, the participant will not remain in the study for further evaluation. See the SoA for data to be collected at the time of discontinuation of study intervention.

## 7.1.1. ECG Changes

A participant who meets either bulleted criterion based on the average of triplicate ECG readings will be withdrawn from the study intervention.

- OTcF >500 msec.
- Change from baseline: QTcF >60 msec and QTcF >450 msec.

If a clinically significant finding is identified (including, but not limited to, changes from baseline in QTcF after enrollment), the investigator or qualified designee will determine if the participant can continue in the study and if any change in participant management is needed. This review of the ECG printed at the time of collection must be documented. Any new clinically relevant finding should be reported as an AE.

## 7.1.2. Potential Cases of Acute Kidney Injury

Abnormal values in SCr concurrent with presence or absence of increase in BUN that meet the criteria below, in the absence of other causes of kidney injury, are considered potential cases of acute kidney injury and should be considered important medical events.

An increase of  $\geq$ 0.3 mg/dL (or  $\geq$ 26.5  $\mu$ mol/L) in SCr level relative to the participant's own baseline measurement should trigger a halt/stopping of dosing, followed by another assessment of SCr as soon as practically feasible, preferably within 48 hours from awareness.

If the second assessment (after the first observations of  $\geq$ 0.3 mg/dL [or  $\geq$ 26.5  $\mu$ mol/L] in SCr relative to the participant's own baseline measurement) confirms the observation of  $\geq$ 0.3 mg/dL (or  $\geq$ 26.5  $\mu$ mol/L), the participant should be discontinued from the study and adequate, immediate, supportive measures taken to correct apparent acute kidney injury.

Participants should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal SCr result. This evaluation should include laboratory tests, detailed history, and physical assessment. In addition to repeating SCr, laboratory tests should include serum BUN, serum creatine kinase, and serum electrolytes (including at a minimum potassium, sodium, phosphate/phosphorus, and calcium), in addition to urinary dipstick, urine microscopic examination, and urinary indices. All cases confirmed on repeat testing as meeting the laboratory criteria for acute kidney injury, with no other cause(s) of laboratory abnormalities identified, should be considered potential cases of drug-induced kidney injury irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal SCr. If  $\geq 2$  healthy participants are noted to have 2 <u>consecutive</u> SCr results change from baseline of  $\geq 0.3$  mg/dL (or  $\geq 26.5$  µmol/L), an assessment of whether the finding may be considered an adverse drug reaction should be undertaken.

#### 7.1.3. Stopping Rules

Dosing will be halted at any time if 1 of the following circumstances occurs and it is determined by the investigator that the occurrence is at least possibly related to the administration of study drug:

- A SAE (eg, a serious AE considered at least possibly related to study drug administration) in 1 participant.
- Severe NSAE (eg, severe NSAEs considered at least possibly related to study drug administration) in 2 participants, independent of within or not within the same SOC.

When stopping rules are met, a data review will be conducted by the sponsor and investigator. If integrated analysis of available data leads to the conclusion that further dosing is justified, an amendment to the protocol may be required if additional safety monitoring is warranted.

## 7.2. Participant Discontinuation/Withdrawal From the Study

A participant may withdraw from the study at any time at his/her own request. Reasons for discontinuation from the study include the following:

- Refused further study procedures;
- Lost to follow-up;
- Death;
- Study terminated by sponsor;
- Investigator's decision
- Pregnancy

At the time of discontinuing from the study, if possible, an early discontinuation visit should be conducted. See the SoA for assessments to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

The early discontinuation visit applies only to participants who are enrolled/randomized and then are prematurely withdrawn from the study. Participants should be questioned regarding their reason for withdrawal.

The participant will be permanently discontinued from the study intervention and the study at that time.

If a participant withdraws from the study, he/she may request destruction of any remaining samples taken and not tested, and the investigator must document any such requests in the site study records and notify the sponsor accordingly.

If the participant withdraws from the study and also withdraws consent (see Section 7.2.1) for disclosure of future information, no further evaluations should be performed and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

#### 7.2.1. Withdrawal of Consent

Participants who request to discontinue receipt of study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact

with him or her or persons previously authorized by the participant to provide this information. Participants should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of study intervention or also from study procedures and/or posttreatment study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

## 7.3. Lost to Follow up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to attend a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible. Counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether the participant wishes to and/or should continue in the study;
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record;
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

The investigator (or an appropriate delegate at the investigator site) must obtain a signed and dated ICD before performing any study-specific procedures.

Study procedures and their timing are summarized in the SoA. Protocol waivers or exemptions are not allowed.

Safety issues should be discussed with the sponsor immediately upon occurrence or awareness to determine whether the participant should continue or discontinue study intervention.

Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

Participants will be screened within 28 days prior to administration of the study intervention to confirm that they meet the study population criteria for the study. If the time between screening and dosing exceeds 28 days as a result of unexpected delays (eg, delayed drug shipment), then participants do not require rescreening if the laboratory results obtained prior to first dose administration meet eligibility criteria.

Every effort should be made to ensure that protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside the control of the investigator that may make it unfeasible to perform the test. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the participant. When a protocol-required test cannot be performed, the investigator will document the reason for the missed test and any corrective and preventive actions that he or she has taken to ensure that required processes are adhered to as soon as possible. The study team must be informed of these incidents in a timely manner.

If an IV catheter is utilized for blood sample collections, ECGs and vital sign assessments (PR and BP) should be collected prior to the insertion of the catheter.

For samples being collected and shipped, detailed collection, processing, storage, and shipment instructions and contact information will be provided to the investigator site prior to initiation of the study.

The total blood sampling volume for individual participants in this study is approximately 260 mL. The actual collection times of blood sampling may change. Additional blood samples may be taken for safety assessments at times specified by Pfizer, provided the total volume taken during the study does not exceed 550 mL during any period of 56 consecutive days.

To prepare for study participation, participants will be instructed on the information in Protocol Section 5.3 Lifestyle Considerations and Section 6.8 Concomitant Therapy.

#### 8.1. Efficacy Assessments

Not applicable.

#### 8.2. Safety Assessments

Planned time points for all safety assessments are provided in the SoA. Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

## 8.2.1. Physical Examinations

A complete PE will include, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems.

A brief physical examination will include, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant-reported symptoms.

Physical examinations may be conducted by a physician, trained physician's assistant, or nurse practitioner as acceptable according to local regulation.

Height and weight will also be measured and recorded as per the SoA. For measuring weight, a scale with appropriate range and resolution is used and must be placed on a stable, flat surface. Participants must remove shoes, bulky layers of clothing, and jackets so that only light clothing remains. They must also remove the contents of their pockets and remain still during measurement of weight.

Physical examination findings collected during the study will be considered source data and will not be required to be reported, unless otherwise noted. Any untoward physical examination findings that are identified during the active collection period and meet the definition of an AE or SAE (Appendix 3) must be reported according to the processes in Sections 8.3.1 to 8.3.3.

#### 8.2.2. Vital Signs

Supine BP will be measured with the participant's arm supported at the level of the heart and recorded to the nearest mm Hg after approximately 5 minutes of rest. The same arm (preferably the dominant arm) will be used throughout the study. Participants should be instructed not to speak during measurements.

The same properly sized and calibrated BP cuff will be used to measure BP each time. The use of an automated device for measuring BP and pulse rate is acceptable; however, when done manually, pulse rate will be measured in the brachial/radial artery for at least 30 seconds. When the timing of these measurements coincides with a blood collection, BP and pulse rate should be obtained prior to the nominal time of the blood collection.

Additional collection times, or changes to collection times, of BP and pulse rate will be permitted, as necessary, to ensure appropriate collection of safety data.

# 8.2.2.1. Respiratory Rate

Respiratory rate will be measured after approximately 5 minutes of rest in a supine position by observing and counting the respirations of the participant for 30 seconds and multiplying by 2. When BP is to be taken at the same time, respiration measurement will be done during the 5 minutes of rest and before BP measurement.

# 8.2.2.2. Temperature

Temperature will be measured orally. No eating, drinking, or smoking is allowed for 15 minutes prior to the measurement.

#### 8.2.3. Electrocardiograms

Standard 12-lead ECGs utilizing limb leads (with a 10 second rhythm strip) should be collected at times specified in the SoA section of this protocol using an ECG machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. Alternative lead placement methodology using torso leads (eg, Mason-Likar) should not be used given the potential risk of discrepancies with ECGs acquired using standard limb lead placement. All scheduled ECGs should be performed after the participant has rested quietly for at least 5 minutes in a supine position.

Triplicate 12-lead ECGs will be obtained approximately 2 minutes apart; the average of the triplicate ECG measurements collected will be recorded.

To ensure safety of the participants, a qualified individual at the investigator site will make comparisons to baseline measurements. Additional ECG monitoring will occur if a) a post dose QTcF interval is increased by ≥60 msec from the baseline **and** is >450 msec; or b) an absolute QT value is ≥500 msec for any scheduled ECG. If either of these conditions occurs, then 2 additional ECGs will be collected approximately 2 to 4 minutes apart to confirm the original measurement. If the QTc values from these repeated ECGs remain above the threshold value, then a single ECG must be repeated at least hourly until QTc values from 2 successive ECGs fall below the threshold value that triggered the repeat measurement.

If a) a post dose QTcF interval remains ≥60 msec from the baseline <u>and</u> is >450 msec; or b) an absolute QT value is ≥500 msec for any scheduled ECG for greater than 4 hours (or sooner, at the discretion of the investigator); or c) QTcF intervals get progressively longer, the participant should undergo continuous ECG monitoring. A cardiologist should be consulted if QTcF intervals do not return to less than the criteria listed above after 8 hours of monitoring (or sooner, at the discretion of the investigator).

In some cases, it may be appropriate to repeat abnormal ECGs to rule out improper lead placement as contributing to the ECG abnormality. It is important that leads be placed in the same positions each time in order to achieve precise ECG recordings. If a machine-read QTc value is prolonged, as defined above, repeat measurements may not be necessary if a qualified medical provider's interpretation determines that the QTcF values are in the acceptable range.

ECG values of potential clinical concern are listed in Appendix 7.

#### 8.2.4. Clinical Safety Laboratory Assessments

See Appendix 2 for the list of clinical safety laboratory tests to be performed and the SoA for the timing and frequency. All protocol-required laboratory assessments, as defined in Appendix 2, must be conducted in accordance with the laboratory manual and the SoA.

Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

The investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.

All laboratory tests with values considered clinically significantly abnormal during participation in the study or within 48 hours after the last dose of study intervention should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the investigator or medical monitor.

If such values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified and the sponsor notified.

See Appendix 6 for suggested actions and follow-up assessments in the event of potential drug-induced liver injury.

## 8.2.5. COVID-19 Specific Assessments

Participants will be tested for SARS-COV-2 infection by PCR prior to being admitted to the CRU for confinement and a subsequent SARS-CoV-2 test will be performed after 4 days (ie, upon completion of  $4 \times 24$  hours in house), or if they develop COVID-19 like symptoms. Additional testing may be required by local regulations or by the Principal Investigator.

## 8.2.6. Pregnancy Testing

Pregnancy tests may be urine or serum tests, but must have a sensitivity of at least 25 mIU/mL. Pregnancy tests will be performed in WOCBP at the times listed in the SoA. Following a negative pregnancy test result at screening, appropriate contraception must be commenced and a second negative pregnancy test result will be required at the baseline visit prior the participant's receiving the study intervention. Pregnancy tests will also be done whenever 1 menstrual cycle is missed during the active treatment period (or when potential pregnancy is otherwise suspected) and at the end of the study. Pregnancy tests may also be repeated if requested by IRBs/ECs or if required by local regulations. If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded if the serum pregnancy result is positive.

#### 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting

The definitions of an AE and an SAE can be found in Appendix 3.

AEs may arise from symptoms or other complaints reported to the investigator by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative), or they may arise from clinical findings of the Investigator or other healthcare providers (clinical signs, test results, etc.).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible to pursue and obtain adequate information both to determine the outcome and to assess whether the event meets the criteria for classification as an SAE or caused the participant to discontinue the study intervention (see Section 7.1).

During the active collection period as described in Section 8.3.1, each participant will be questioned about the occurrence of AEs in a nonleading manner.

In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion.

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant begins from the time the participant provides informed consent, which is obtained before the participant's participation in the study (ie, before undergoing any study-related procedure and/or receiving study intervention), through and including a minimum of 28 calendar days, except as indicated below, after the last administration of the study intervention.

Follow-up by the investigator continues throughout and after the active collection period and until the AE or SAE or its sequelae resolve or stabilize at a level acceptable to the investigator.

For participants who are screen failures, the active collection period ends when screen failure status is determined.

If the participant withdraws from the study and also withdraws consent for the collection of future information, the active collection period ends when consent is withdrawn.

If a participant permanently discontinues or temporarily discontinues study intervention because of an AE or SAE, the AE or SAE must be recorded on the CRF and the SAE reported using the CT SAE Report Form.

Investigators are not obligated to actively seek information on AEs or SAEs after the participant has concluded study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has completed the study, and he/she considers the event to be reasonably related to the study intervention, the investigator must promptly report the SAE to Pfizer using the CT SAE Report Form.

# 8.3.1.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a participant during the active collection period as described in Section 8.3.1 are reported to Pfizer Safety on the CT SAE Report Form immediately upon awareness and under no circumstance should this exceed 24 hours, as indicated in

Appendix 3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

## 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF

All nonserious AEs and SAEs occurring in a participant during the active collection period, which begins after obtaining informed consent as described in Section 8.3.1, will be recorded on the AE section of the CRF.

The investigator is to record on the CRF all directly observed and all spontaneously reported AEs and SAEs reported by the participant.

#### 8.3.2. Method of Detecting AEs and SAEs

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

#### 8.3.3. Follow-Up of AEs and SAEs

After the initial AE or SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. For each event, the investigator must pursue and obtain adequate information until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3).

In general, follow-up information will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a participant death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety.

Further information on follow-up procedures is given in Appendix 3.

## 8.3.4. Regulatory Reporting Requirements for SAEs

Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities toward the safety of participants and the safety of a study intervention under clinical investigation are met.

The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ECs, and investigators.

Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

An investigator who receives SUSARs or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the SRSD(s) for the study and will notify the IRB/EC, if appropriate according to local requirements.

# 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure

Environmental exposure occurs when a person not enrolled in the study as a participant receives unplanned direct contact with or exposure to the study intervention. Such exposure may or may not lead to the occurrence of an AE or SAE. Persons at risk for environmental exposure include healthcare providers, family members, and others who may be exposed. An environmental exposure may include exposure during pregnancy, exposure during breastfeeding, and occupational exposure.

Any such exposure to the study intervention under study are reportable to Pfizer Safety within 24 hours of investigator awareness.

## 8.3.5.1. Exposure During Pregnancy

An EDP occurs if:

- A female participant is found to be pregnant while receiving or after discontinuing study intervention.
- A male participant who is receiving or has discontinued study intervention exposes a female partner prior to or around the time of conception.
- A female is found to be pregnant while being exposed or having been exposed to study intervention due to environmental exposure. Below are examples of environmental EDP:
  - A female family member or healthcare provider reports that she is pregnant after having been exposed to the study intervention by ingestion, inhalation, or skin contact.
  - A male family member or healthcare provider who has been exposed to the study intervention by ingestion, inhalation, or skin contact then exposes his female partner prior to or around the time of conception.

The investigator must report EDP to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The initial information submitted

should include the anticipated date of delivery (see below for information related to termination of pregnancy).

- If EDP occurs in a participant or a participant's partner, the investigator must report this information to Pfizer Safety on the CT SAE Report Form and an EDP Supplemental Form, regardless of whether an SAE has occurred. Details of the pregnancy will be collected after the start of study intervention and until 28 days after the last dose.
- If EDP occurs in the setting of environmental exposure, the investigator must report information to Pfizer Safety using the CT SAE Report Form and EDP Supplemental Form. Since the exposure information does not pertain to the participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed CT SAE Report Form is maintained in the investigator site file.

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP Supplemental Form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless preprocedure test findings are conclusive for a congenital anomaly and the findings are reported).

Abnormal pregnancy outcomes are considered SAEs. If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly in a live-born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death), the investigator should follow the procedures for reporting SAEs. Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion including miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the study intervention.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the participant with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the participant was given the Pregnant Partner Release of Information Form to provide to his partner.

## 8.3.5.2. Exposure During Breastfeeding

An exposure during breastfeeding occurs if:

- A female participant is found to be breastfeeding while receiving or after discontinuing study intervention.
- A female is found to be breastfeeding while being exposed or having been exposed to study intervention (ie, environmental exposure). An example of environmental exposure during breastfeeding is a female family member or healthcare provider who reports that she is breastfeeding after having been exposed to the study intervention by ingestion, inhalation, or skin contact.

The investigator must report exposure during breastfeeding to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The information must be reported using the CT SAE Report Form. When exposure during breastfeeding occurs in the setting of environmental exposure, the exposure information does not pertain to the participant enrolled in the study, so the information is not recorded on a CRF. However, a copy of the completed CT SAE Report Form is maintained in the investigator site file.

An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug, the SAE is reported together with the exposure during breastfeeding.

# 8.3.5.3. Occupational Exposure

The investigator must report any instance of occupational exposure to Pfizer Safety within 24 hours of the investigator's awareness using the CT SAE Report Form regardless of whether there is an associated SAE. Since the information about the occupational exposure does not pertain to a participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed CT SAE Report Form must be maintained in the investigator site file.

#### 8.3.6. Cardiovascular and Death Events

Not applicable.

# 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs

Not applicable.

## 8.3.8. Adverse Events of Special Interest

Adverse events of special interest (AESIs) are examined as part of routine safety data review procedures throughout the clinical trial and as part of signal detection processes.

All AESIs must be reported as an AE or SAE following the procedures described in Section 8.3.1 through 8.3.4. An AESI is to be recorded as an AE or SAE on the CRF. In addition, an AESI that is also an SAE must be reported using the CT SAE Report Form.

## 8.3.8.1. Lack of Efficacy

This section is not applicable because efficacy is not expected in the study population.

#### 8.3.9. Medical Device Deficiencies

Not applicable.

#### 8.3.10. Medication Errors

Medication errors may result from the administration or consumption of the study intervention by the wrong participant, or at the wrong time, or at the wrong dosage strength.

Exposures to the study intervention under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the CT SAE Report<br>Form to Pfizer Safety Within<br>24 Hours of Awareness |
|---|---|---|
| Medication errors | All (regardless of whether associated with an AE) | Only if associated with an SAE |

#### Medication errors include:

- Medication errors involving participant exposure to the study intervention;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the study participant.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified within 24 hours.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and nonserious, are recorded on the AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a CT SAE Report Form **only when associated with an SAE.** 

#### 8.4. Pharmacokinetics

# 8.4.1. Plasma for Analysis of PF-07321332 CCI

Blood samples of approximately 4 mL, to provide approximately 1.5 mL plasma, will be collected for measurement of plasma concentrations of PF-07321332 as specified in the SoA. Instructions for the collection and handling of biological samples will be provided in the laboratory manual or by the sponsor. The actual date and time (24-hour clock time) of each sample will be recorded.

The actual times may change, but the number of samples will remain the same. All efforts will be made to obtain the samples at the exact nominal time relative to dosing. Collection of samples up to and including 10 hours after dose administration that are obtained within 10% of the nominal time relative to dosing (eg, within 6 minutes of a 60-minute sample) will not be captured as a protocol deviation, as long as the exact time of the collection is noted on the source document and the CRF. Collection of samples more than 10 hours after dose administration that are obtained ≤1 hour away from the nominal time relative to dosing will not be captured as a protocol deviation, as long as the exact time of the collection is noted on the source document and the CRF.

Samples will be used to evaluate the PK of PF-07321332 CCI . Samples collected for analyses of PF-07321332 concentration may also be used to evaluate safety or efficacy aspects related to concerns arising during or after the study, for metabolite identification, analysis of endogenous biomarkers, and/or evaluation of the bioanalytical method, CCI

Genetic analyses will not be performed on these plasma samples unless consent for this was included in the informed consent. Participant confidentiality will be maintained.

Samples collected for measurement of plasma concentrations of PF-07321332 will be analyzed using a validated analytical method in compliance with applicable SOPs. Potential metabolites may be analyzed with either validated methods.

The PK samples must be processed and shipped as indicated in the instructions provided to the investigator site to maintain sample integrity. Any deviations from the PK sample handling procedure (eg, sample collection and processing steps, interim storage or shipping conditions), including any actions taken, must be documented and reported to the sponsor. On a case-by-case basis, the sponsor may make a determination as to whether sample integrity has been compromised.

Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/EC will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the ICD.

## 8.5. Genetics

# 8.5.1. Specified Genetics

Genetics (specified analyses) are not evaluated in this study.



#### 8.6. Biomarkers

Biomarkers are not evaluated in this study.

## 8.6.1. Specified Gene Expression (RNA) Research

Specified gene expression (RNA) research is not included in this study.

# **8.6.2. Specified Protein Research**

Specified protein research is not included in this study.

## 8.6.3. Specified Metabolomic Research

Specified metabolomic research is not included in this study.



## 8.7. Immunogenicity Assessments

Immunogenicity assessments are not included in this study.

#### 8.8. Health Economics

Health economics/medical resource utilization and health economics parameters are not evaluated in this study.

#### 9. STATISTICAL CONSIDERATIONS

Detailed methodology for summary and statistical analyses of the data collected in this study is outlined here and further detailed in a SAP, which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

# 9.1. Statistical Hypotheses

There are no statistical hypotheses for this study.

## 9.2. Analysis Sets

For purposes of analysis, the following analysis sets are defined:

| Participant Analysis<br>Set | Description |
|---|---|
| Enrolled/Randomly assigned to study intervention | "Enrolled" means a participant's, or their legally authorized representative's, agreement to participate in a clinical study following completion of the informed consent process and screening. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening. |
| Safety Analysis Set | All participants who take at least 1 dose of study intervention. Participants will be analyzed according to the product they actually received. |
| PK Concentration Set | All participants who take at least 1 dose of study intervention and in whom at least 1 concentration value is reported. |
| PK Parameter Set | All participants who take at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest are reported. |

## 9.3. Statistical Analyses

The SAP will be developed and finalized before any analyses are performed and will describe the analyses and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary and secondary endpoints.

## 9.3.1. Pharmacokinetic Analyses

#### 9.3.1.1. Derivation of Pharmacokinetic Parameters

Plasma PK parameters of PF-07321332 will be derived (as data permit) from the concentration-time data using standard noncompartmental methods as outlined in the Table below. Actual PK sampling times will be used in the derivation of PK parameters. In the case that actual PK sampling times are not available, nominal PK sampling time will be used in the derivation of PK parameters.

Plasma PF-07321332 CCI PK Parameters Definitions

| Parameter | Definition | Method of Determination |
|---|---|---|
| AUC <sub>last</sub> | Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (C <sub>last</sub> ). | Linear/Log trapezoidal method. |
| AUC <sub>tau</sub> | Area under the plasma concentration-time profile from time zero to time tau $(\tau)$ , where tau=12-hour dosing interval. | Linear/Log trapezoidal method. |
| $C_{max}$ | Maximum observed concentration | Observed directly from data |
| T <sub>max</sub> | Time for C <sub>max</sub> | Observed directly from data as time of first occurrence |
| t <sub>1/2</sub> * | Terminal half-life | Log <sub>e</sub> (2)/k <sub>el</sub> , where k <sub>el</sub> is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. Only those data points judged to describe the terminal loglinear decline will be used in the regression. |
| CL/F | Apparent clearance | Dose/AUC <sub>tau</sub> |
| V <sub>z</sub> /F* | Apparent volume of distribution | Dose/(AUC <sub>tau</sub> • k <sub>el</sub> ) |

<sup>\*</sup>If data permit.

#### 9.3.2. Statistical Methods for PK Data

The plasma concentrations of PF-07321332 CCI will be listed and descriptively summarized by nominal PK sampling time and treatment. Individual participant, as well as mean and median profiles of the plasma concentration time data will be plotted by treatment for each analyte using actual (for individual) and nominal (for mean and median) times respectively. Mean and median profiles will be presented on both linear and semi-log scales. Box and whisker plots for AUC<sub>tau</sub> and C<sub>max</sub> following multiple doses of PF-07321332/ritonavir will be plotted by treatment.

Natural log transformed parameters (AUC<sub>tau</sub>, and C<sub>max</sub>) of PF-07321332 will be analyzed using a mixed effect model with treatment as fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs will be obtained from the model. The adjusted mean differences and 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. PF-07321332/ritonavir administered alone will be the Reference treatment and PF-07321332/ritonavir co-administered with itraconazole will be the Test treatment.

Additional specifications about the tables, listings, and figures will be outlined in the SAP.

## 9.3.3. Other Safety Analyses

All safety analyses will be performed on the safety population.

AEs, ECGs, BP, PR, and safety laboratory data will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of participants. Any clinical laboratory, ECG, BP, and PR abnormalities of potential clinical concern will be described. Safety data will be presented in tabular and/or graphical format and summarized descriptively, where appropriate.

Medical history and PE and neurological examination information, as applicable, collected during the course of the study will be considered source data and will not be required to be reported, unless otherwise noted. However, any untoward findings identified on physical and/or neurological examinations conducted during the active collection period will be captured as AEs, if those findings meet the definition of an AE. Data collected at Screening that are used for inclusion/exclusion criteria, such as laboratory data, ECGs, and vital signs, will be considered source data, and will not be required to be reported, unless otherwise noted. Demographic data collected at Screening will be reported.



## 9.4. Interim Analyses

No formal interim analysis will be conducted for this study. As this is an open-label study, the sponsor may conduct unblinded reviews of the data during the course of the study for the purpose of safety assessment, facilitating PK/PD modeling, and/or supporting clinical development.

## 9.5. Sample Size Determination

A sample size of 9 participants will provide adequate precision to estimate the effects of itraconazole on the PK of PF-07321332. The expected widths of the 90% CIs with 80% coverage probability are shown in the following table for a range of possible effects.

| Parameter | Estimated Effect (100*Test/Reference) | 90% CI | CI Width |
|-------------|---------------------------------------|------------|----------|
| $AUC_{tau}$ | 100% | 88%, 113% | 25% |
| | 110% | 97%, 124% | 27% |
| | 120% | 106%, 136% | 30% |
| | 130% | 115%, 147% | 32% |
| | 140% | 124%, 158% | 35% |
| $C_{max}$ | 100% | 92%, 108% | 16% |
| | 110% | 102%, 119% | 17% |
| | 120% | 111%, 130% | 19% |
| | 130% | 120%, 141% | 21% |
| | 140% | 129%, 152% | 22% |

These estimates are based on the assumption that within-participant standard deviations are 0.14 and 0.091 for  $lnAUC_{tau}$  and  $lnC_{max}$ , respectively, as obtained from ongoing clinical study C4671001 in healthy participants.

To allow for dropouts, 12 participants will be enrolled in order to have 9 PK evaluable participants. Participants who withdraw from the study may be replaced at the discretion of the investigator upon consultation with the sponsor.

#### 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1. Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and CIOMS International Ethical Guidelines;
- Applicable ICH GCP guidelines;
- Applicable laws and regulations, including applicable privacy laws.

The protocol, protocol amendments, ICD, SRSD(s), and other relevant documents (eg, advertisements) must be reviewed and approved by the sponsor, submitted to an IRB/EC by the investigator, and reviewed and approved by the IRB/EC before the study is initiated.

Any amendments to the protocol will require IRB/EC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

Protocols and any substantial amendments to the protocol will require health authority approval prior to initiation except for changes necessary to eliminate an immediate hazard to study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC;
- Notifying the IRB/EC of SAEs or other significant safety findings as required by IRB/EC procedures;
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH GCP guidelines, the IRB/EC, European regulation 536/2014 for clinical studies (if applicable), European Medical Device Regulation 2017/745 for clinical device research (if applicable), and all other applicable local regulations.

# 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the study intervention, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study participants against any immediate hazard, and of any serious breaches of this protocol or of the ICH GCP guidelines that the investigator becomes aware of.

#### 10.1.2. Informed Consent Process

The investigator or his/her representative will explain the nature of the study, including the risks and benefits, to the participant and answer all questions regarding the study. The participant should be given sufficient time and opportunity to ask questions and to decide whether or not to participate in the trial.

Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, privacy and data protection requirements, where applicable, and the IRB/EC or study center.

The investigator must ensure that each study participant is fully informed about the nature and objectives of the study, the sharing of data related to the study, and possible risks associated with participation, including the risks associated with the processing of the participant's personal data.

The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.

The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/EC members, and by inspectors from regulatory authorities.

The investigator further must ensure that each study participant is fully informed about his or her right to access and correct his or her personal data and to withdraw consent for the processing of his or her personal data.

The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date on which the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICD.

Participants must be reconsented to the most current version of the ICD(s) during their participation in the study.

A copy of the ICD(s) must be provided to the participant.

A participant who is rescreened is not required to sign another ICD if the rescreening occurs within 10 days from the previous ICD signature date.

#### 10.1.3. Data Protection

All parties will comply with all applicable laws, including laws regarding the implementation of organizational and technical measures to ensure protection of participant data.

Participants' personal data will be stored at the study site in encrypted electronic and/or paper form and will be password-protected or secured in a locked room to ensure that only authorized study staff have access. The study site will implement appropriate technical and organizational measures to ensure that the personal data can be recovered in the event of disaster. In the event of a potential personal data breach, the study site will be responsible for determining whether a personal data breach has in fact occurred and, if so, providing breach notifications as required by law.

To protect the rights and freedoms of participants with regard to the processing of personal data, participants will be assigned a single, participant-specific numerical code. Any participant records or data sets that are transferred to the sponsor will contain the numerical code; participant names will not be transferred. All other identifiable data transferred to the sponsor will be identified by this single, participant-specific code. The study site will maintain a confidential list of participants who participated in the study, linking each participant's numerical code to his or her actual identity and medical record ID. In case of data transfer, the sponsor will protect the confidentiality of participants' personal data consistent with the clinical study agreement and applicable privacy laws.

#### 10.1.4. Committees Structure

#### 10.1.4.1. Data Monitoring Committee

This study will not use a DMC.

## 10.1.5. Dissemination of Clinical Study Data

Pfizer fulfills its commitment to publicly disclose clinical study results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the EudraCT, and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations. In addition, Pfizer reports study results outside of the requirements of local laws/regulations pursuant to its SOPs.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

## www.clinicaltrials.gov

Pfizer posts clinical trial results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a product, regardless of the geographical location in which the study is conducted. These results are submitted for posting in accordance with the format and timelines set forth by US law.

#### **EudraCT**

Pfizer posts clinical trial results on EudraCT for Pfizer-sponsored interventional studies in accordance with the format and timelines set forth by EU requirements.

## www.pfizer.com

Pfizer posts public disclosure synopses (CSR synopses in which any data that could be used to identify individual participants have been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the corresponding study results are posted to www.clinicaltrials.gov.

## Documents within marketing authorization packages/submissions

Pfizer complies with the European Union Policy 0070, the proactive publication of clinical data to the EMA website. Clinical data, under Phase 1 of this policy, includes clinical overviews, clinical summaries, CSRs, and appendices containing the protocol and protocol amendments, sample CRFs, and statistical methods. Clinical data, under Phase 2 of this policy, includes the publishing of individual participant data. Policy 0070 applies to new marketing authorization applications submitted via the centralized procedure since 01 January 2015 and applications for line extensions and for new indications submitted via the centralized procedure since 01 July 2015.

## Data sharing

Pfizer provides researchers secure access to patient-level data or full CSRs for the purposes of "bona-fide scientific research" that contributes to the scientific understanding of the disease, target, or compound class. Pfizer will make data from these trials available 24 months after study completion. Patient-level data will be anonymized in accordance with applicable privacy laws and regulations. CSRs will have personally identifiable information redacted.

Data requests are considered from qualified researchers with the appropriate competencies to perform the proposed analyses. Research teams must include a biostatistician. Data will not be provided to applicants with significant conflicts of interest, including individuals requesting access for commercial/competitive or legal purposes.

#### **10.1.6.** Data Quality Assurance

All participant data relating to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

Guidance on completion of CRFs will be provided in the CRF Completion Requirements document.

The investigator must ensure that the CRFs are securely stored at the study site in encrypted electronic and/or paper form and are password-protected or secured in a locked room to prevent access by unauthorized third parties.

The investigator must permit study-related monitoring, audits, IRB/EC review, and regulatory agency inspections and provide direct access to source data documents. This verification may also occur after study completion. It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

Monitoring details describing strategy, including definition of study critical data items and processes (eg, risk-based initiatives in operations and quality, such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, virtual, or on-site monitoring), are provided in the IQMP.

The sponsor or designee is responsible for the data management of this study, including quality checking of the data.

Records and documents, including signed ICDs, pertaining to the conduct of this study must be retained by the investigator for 15 years after study completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor. The investigator must ensure that the records continue to be stored securely for as long as they are maintained.

When participant data are to be deleted, the investigator will ensure that all copies of such data are promptly and irrevocably deleted from all systems.

The investigator(s) will notify the sponsor or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with the sponsor or its agents to prepare the investigator site for the inspection and will allow the sponsor or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the participant's medical records. The investigator will promptly provide copies of the inspection findings to the sponsor or its agent. Before response submission to the regulatory authorities, the investigator will provide the sponsor or its agents with an opportunity to review and comment on responses to any such findings.

#### 10.1.7. Source Documents

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator site.

Data reported on the CRF or entered in the eCRF that are from source documents must be consistent with the source documents or the discrepancies must be explained. The

investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Definition of what constitutes source data and its origin can be found the Source Document Locator, which is maintained by the sponsor's designee (Pfizer Clinical Research Unit).

Description of the use of the computerized system is documented in the Source Document Locator, which is maintained by the sponsor's designee (Pfizer Clinical Research Unit).

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP guidelines, and all applicable regulatory requirements.

## 10.1.8. Study and Site Start and Closure

The study start date is the date on which the clinical study will be open for recruitment of participants.

The first act of recruitment is the date of the first participant's first visit and will be the study start date.

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time upon notification to the sponsor if requested to do so by the responsible IRB/EC or if such termination is required to protect the health of study participants.

Reasons for the early closure of a study site by the sponsor may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/EC or local health authorities, the sponsor's procedures, or the ICH GCP guidelines;
- Inadequate recruitment of participants by the investigator;
- Discontinuation of further study intervention development.

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the ECs/IRBs, the regulatory authorities, and any CRO(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

Study termination is also provided for in the clinical study agreement. If there is any conflict between the contract and this protocol, the contract will control as to termination rights.

## 10.1.9. Publication Policy

The results of this study may be published or presented at scientific meetings by the investigator after publication of the overall study results or 1 year after the end of the study (or study termination), whichever comes first.

The investigator agrees to refer to the primary publication in any subsequent publications, such as secondary manuscripts, and submits all manuscripts or abstracts to the sponsor 30 days before submission. This allows the sponsor to protect proprietary information and to provide comments, and the investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer-intervention related information necessary for the appropriate scientific presentation or understanding of the study results.

For all publications relating to the study, the investigator will comply with recognized ethical standards concerning publications and authorship, including those established by the International Committee of Medical Journal Editors.

The sponsor will comply with the requirements for publication of the overall study results covering all investigator sites. In accordance with standard editorial and ethical practice, the sponsor will support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship of publications for the overall study results will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

If publication is addressed in the clinical study agreement, the publication policy set out in this section will not apply.

## 10.1.10. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in CTMS

To facilitate access to appropriately qualified medical personnel for study-related medical questions or problems, participants are provided with an Emergency Contact Card (ECC) at

the time of informed consent. The ECC contains, at a minimum, (a) protocol and study intervention identifiers, (b) participant's study identification number, (c) site emergency phone number active 24 hours/day, 7 days per week.

The ECC is intended to augment, not replace, the established communication pathways between the investigator, site staff, and study team. The ECC is to be used by healthcare professionals not involved in the research study only, as a means of reaching the investigator or site staff related to the care of a participant.

## 10.2. Appendix 2: Clinical Laboratory Tests

The following safety laboratory tests will be performed at times defined in the SoA section of this protocol. Additional laboratory results may be reported on these samples as a result of the method of analysis or the type of analyzer used by the clinical laboratory, or as derived from calculated values. These additional tests would not require additional collection of blood. Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

| Table 1. | Protocol | -Required S | Safety | Laboratory | Assessments | • |
|----------|----------|-------------|--------|------------|-------------|---|
| | | | | | | _ |

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hemoglobin | BUN and creatinine | Local Dipstick: | • SARS-CoV-2 RT-PCR |
| Hematocrit | Glucose (fasting) | pН | Urine drug screening <sup>c</sup> |
| RBC count | Calcium | Glucose (qual) | <ul> <li>Pregnancy test (β-hCG)<sup>d</sup></li> </ul> |
| MCV | Sodium | Protein (qual) | • eGFR [CKD-EPI] |
| MCH | Potassium | Blood (qual) | • aPTT |
| MCHC | Chloride | Ketones | PT-INR |
| Platelet count | Total CO <sub>2</sub> (bicarbonate) | Nitrites | • Fibrinogen |
| WBC count | AST, ALT | Leukocyte esterase | • CCI |
| Total neutrophils (Abs) | Total bilirubin | | |
| Eosinophils (Abs) | Alkaline phosphatase | <u>Laboratory:</u> | |
| Monocytes (Abs) Basophils (Abs) Lymphocytes (Abs) | Uric acid Albumin Total protein | Microscopy and<br>Culture <sup>a</sup> | At Screening only: FSH <sup>b</sup> HBsAg HBsAb HBcAb HCVAb |

- a. Only if urine dipstick is positive for blood, protein, nitrites, or leukocyte esterase and culture only if bacteriuria.
- b. For confirmation of postmenopausal status only.
- c. At screening and Day -1; The minimum requirement for drug screening includes cocaine, THC, opiates/opioids, benzodiazepines, and amphetamines (others are site and study specific).
- d. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/EC. Serum or urine β-hCG for female participants of childbearing potential.

The investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF.

Any remaining serum/plasma from samples collected for clinical safety laboratory measurements at baseline and at all times after dose administration may be retained and stored for the duration of the study.

These data will not be included in the CSR. Samples to be used for this purpose will be shipped to either a Pfizer-approved BBS facility or other designated laboratory and retained for up to 1 year following the completion of the study.

# 10.3. Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting

#### 10.3.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

## **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (eg, ECG, radiological scans, vital sign measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator. Any abnormal laboratory test results that meet any of the conditions below must be recorded as an AE:
  - Is associated with accompanying symptoms;
  - Requires additional diagnostic testing or medical/surgical intervention;
  - Leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
- Exacerbation of a chronic or intermittent preexisting condition, including either an increase in frequency and/or intensity of the condition.
- New condition detected or diagnosed after study intervention administration, even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE or SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

## **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2. Definition of an SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed below:

#### a. Results in death

#### b. Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

# c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a preexisting condition that did not worsen from baseline is not considered an AE.

## d. Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance, such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle), that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

# e. Is a congenital anomaly/birth defect

# f. Is a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, is considered serious.

The event may be suspected from clinical symptoms or laboratory findings indicating an infection in a participant exposed to a Pfizer product. The terms "suspected transmission" and "transmission" are considered synonymous. These cases are considered unexpected and handled as serious expedited cases by pharmacovigilance personnel. Such cases are also considered for reporting as product defects, if appropriate.

#### g. Other situations:

- Medical or scientific judgment should be exercised by the investigator in deciding whether SAE reporting is appropriate in other situations, such as significant medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

# 10.3.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period

#### AE and SAE Recording/Reporting

The table below summarizes the requirements for recording AEs on the CRF and for reporting SAEs on the CT SAE Report Form to Pfizer Safety throughout the active collection period. These requirements are delineated for 3 types of events: (1) SAEs; (2) nonserious AEs; and (3) exposure to the study intervention under study during pregnancy or breastfeeding, and occupational exposure.

It should be noted that the CT SAE Report Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the CT SAE Report Form for reporting of SAE information.

| Safety Event | Recorded on the CRF | Reported on the CT SAE<br>Report Form to Pfizer<br>Safety Within 24 Hours<br>of Awareness |
|---|---|---|
| SAE | All | All |
| Nonserious AE | All | None |
| Exposure to the study intervention under study during pregnancy or breastfeeding | All AEs/SAEs associated with exposure during pregnancy or breastfeeding | All instances of EDP are reported (whether or not there is an associated SAE)* |
| J | <b>Note:</b> Instances of EDP or EDB not associated with an AE or SAE are not captured in the CRF. | All instances of EDB are reported (whether or not there is an associated SAE). ** |
| Environmental or occupational exposure to the product under study to a non-participant (not involving EDP or EDB). | None. Exposure to a study non-participant is not collected on the CRF. | The exposure (whether or not there is an associated AE or SAE) must be reported.*** |

- \* EDP (with or without an associated AE or SAE): any pregnancy information is reported to Pfizer Safety using CT SAE Report Form and EDP Supplemental Form; if the EDP is associated with an SAE, then the SAE is reported to Pfizer Safety using the CT SAE Report Form.
- \*\* **EDB** is reported to Pfizer Safety using the CT SAE Report Form which would also include details of any SAE that might be associated with the EDB.
- \*\*\* Environmental or Occupational exposure: AEs or SAEs associated with occupational exposure are reported to Pfizer Safety using the CT SAE Report Form.
- When an AE or SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.
- The investigator will then record all relevant AE or SAE information in the CRF.

- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of completion of the CT SAE Report Form/AE or SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE or SAE.

## **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to 1 of the following categories:

- Mild: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Moderate: Minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL. Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- Severe: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling, limiting self care ADL. Self care ADL refers to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

An event is defined as "serious" when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

## **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.

- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration, will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has
  minimal information to include in the initial report to the sponsor. However, it is
  very important that the investigator always make an assessment of causality
  for every event before the initial transmission of the SAE data to the
  sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.
- If the investigator does not know whether or not the study intervention caused the event, then the event will be handled as "related to study intervention" for reporting purposes, as defined by the sponsor. In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the CT SAE Report Form and in accordance with the SAE reporting requirements.

#### Follow-Up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations, as medically indicated or as requested by the sponsor, to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide Pfizer Safety with a copy of any postmortem findings, including histopathology.
- New or updated information will be recorded in the originally submitted documents.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 10.3.4. Reporting of SAEs

### SAE Reporting to Pfizer Safety via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to Pfizer Safety will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as the data become available.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section) or to Pfizer Safety by telephone.

#### SAE Reporting to Pfizer Safety via CT SAE Report Form

- Facsimile transmission of the CT SAE Report Form is the preferred method to transmit this information to Pfizer Safety.
- In circumstances when the facsimile is not working, notification by telephone is acceptable with a copy of the CT SAE Report Form sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the CT SAE Report Form pages within the designated reporting time frames.

#### 10.4. Appendix 4: Contraceptive and Barrier Guidance

## 10.4.1. Male Participant Reproductive Inclusion Criteria

Male participants are eligible to participate if they agree to the following requirements during the intervention period and for at least 28 days after the last dose of study intervention, which corresponds to the time needed to eliminate reproductive safety risk of the study intervention(s):

• Refrain from donating sperm.

#### PLUS either:

 Be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

OR

- Must agree to use contraception/barrier as detailed below:
  - Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
- In addition to male condom use, a highly effective method of contraception may be considered in WOCBP partners of male participants (refer to the list of highly effective methods below in Section 10.4.4).

#### 10.4.2. Female Participant Reproductive Inclusion Criteria

A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

• Is not a WOCBP (see definitions below in Section 10.4.3).

OR

• Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, as described below during the intervention period and for at least 28 days after the last dose of study intervention, which corresponds to the time needed to eliminate any reproductive safety risk of the study intervention(s). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

A WOCBP agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

#### 10.4.3. Woman of Childbearing Potential

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (eg, amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before the first dose of study intervention, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- 1. Premenopausal female with 1 of the following:
  - Documented hysterectomy;
  - Documented bilateral salpingectomy;
  - Documented bilateral oophorectomy.

For individuals with permanent infertility due to an alternate medical cause other than the above, (eg, mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

Note: Documentation for any of the above categories can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview. The method of documentation should be recorded in the participant's medical record for the study.

- 2. Postmenopausal female.
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In addition:
    - A high FSH level in the postmenopausal range must be used to confirm a postmenopausal state in women under 60 years old and not using hormonal contraception or HRT.
    - A female on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods

if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### 10.4.4. Contraception Methods

Contraceptive use by men or women should be consistent with local availability/regulations regarding the use of contraceptive methods for those participating in clinical trials.

#### **Highly Effective Methods That Have Low User Dependency**

- 1. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.
- 2. Intrauterine device.
- 3. Intrauterine hormone-releasing system.
- 4. Bilateral tubal occlusion (eg, bilateral tubal ligation).
- 5. Vasectomized partner.
  - A vasectomized partner is a highly effective contraceptive method provided that the partner is the sole sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used. The spermatogenesis cycle is approximately 90 days.



# 10.6. Appendix 6: Liver Safety: Suggested Actions and Follow-Up Assessments Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver enzyme elevations but adapt are termed "adaptors." In some participants, transaminase elevations are a harbinger of a more serious potential outcome. Participants who experience a transaminase elevation above 3 × ULN should be monitored more frequently to determine if they are "adaptors" or are "susceptible."

Abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below need to be evaluated for causality and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities depends on the participant's individual baseline values and underlying conditions. Participants who present with the following laboratory abnormalities should halt/stop dosing and be evaluated for causality to definitively determine the etiology of the abnormal laboratory values:

- Participants with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available.
- For participants with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).
  - Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The participant should return to the investigator site and be evaluated for causality as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment. If on further evaluation the abnormal test result is repeated, the participant should be discontinued from the study and adequate, immediate, supportive measures taken.

In addition to repeating measurements of AST and ALT and TBili for suspected liver toxicity additional laboratory tests should include albumin, CK, direct and indirect bilirubin, GGT, PT/INR, total bile acids, and alkaline phosphatase. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen/paracetamol (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, or supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection, liver imaging (eg, biliary tract), and collection of serum samples for acetaminophen/paracetamol drug and/or protein adduct levels may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI cases if no other reason for the LT abnormalities has yet been found. Such potential DILI cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

#### 10.7. Appendix 7: ECG Findings of Potential Clinical Concern

#### ECG Findings That May Qualify as AEs

- Marked sinus bradycardia (rate <40 bpm) lasting minutes.
- New PR interval prolongation >280 msec.
- New prolongation of QTcF to >480 msec (absolute) or by ≥60 msec from baseline.
- New-onset atrial flutter or fibrillation, with controlled ventricular response rate: ie, rate <120 bpm.
- New-onset type I second-degree (Wenckebach) AV block of >30 seconds' duration.
- Frequent PVCs, triplets, or short intervals (<30 seconds) of consecutive ventricular complexes.

#### ECG Findings That May Qualify as SAEs

- QTcF prolongation >500 msec.
- New ST-T changes suggestive of myocardial ischemia.
- New-onset left bundle branch block (QRS > 120 msec).
- New-onset right bundle branch block (QRS >120 msec).
- Symptomatic bradycardia.
- Asystole:
  - In awake, symptom-free participants in sinus rhythm, with documented periods of asystole ≥3.0 seconds or any escape rate <40 bpm, or with an escape rhythm that is below the AV node.
  - In awake, symptom-free participants with atrial fibrillation and bradycardia with 1 or more pauses of at least 5 seconds or longer.
  - Atrial flutter or fibrillation, with rapid ventricular response rate: rapid = rate >120 bpm.
- Sustained supraventricular tachycardia (rate >120 bpm) ("sustained" = short duration with relevant symptoms or lasting >1 minute).

- Ventricular rhythms >30 seconds' duration, including idioventricular rhythm (heart rate <40 bpm), accelerated idioventricular rhythm (HR >40 bpm to <100 bpm), and monomorphic/polymorphic ventricular tachycardia (HR >100 bpm (such as torsades de pointes)).
- Type II second-degree (Mobitz II) AV block.
- Complete (third-degree) heart block.

#### ECG Findings That Qualify as SAEs

- Change in pattern suggestive of new myocardial infarction.
- Sustained ventricular tachyarrhythmias (>30 seconds' duration).
- Second- or third-degree AV block requiring pacemaker placement.
- Asystolic pauses requiring pacemaker placement.
- Atrial flutter or fibrillation with rapid ventricular response requiring cardioversion.
- Ventricular fibrillation/flutter.
- At the discretion of the investigator, any arrhythmia classified as an adverse experience.

The enumerated list of major events of potential clinical concern are recommended as "alerts" or notifications from the core ECG laboratory to the investigator and Pfizer study team, and not to be considered as all inclusive of what to be reported as AEs/SAEs.

# 10.8. Appendix 8: Abbreviations

The following is a list of abbreviations that may be used in the protocol.

| Abbreviation | Term |
|---|---|
| $\rightarrow$ | ongoing/continuous event |
| 3CL | 3C-like |
| 3CL <sup>pro</sup> | 3C-like protein |
| Abs | absolute |
| ADL | activities of daily living |
| AE | adverse event |
| AESI | adverse events of special interest |
| ALT | alanine aminotransferase |
| aPTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| AUC <sub>last</sub> | area under the plasma concentration-time curve from time 0 to the |
| | time of the last measurable concentration |
| AUC <sub>tau</sub> | area under the plasma concentration-time curve over dosing |
| | interval |
| AV | atrioventricular |
| BBS | Biospecimen Banking System |
| β-hCG | beta-human chorionic gonadotropin |
| BID | twice a day |
| BMI | body mass index |
| BP | blood pressure |
| bpm | beats per minute |
| BUN | blood urea nitrogen |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK | creatine kinase |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| CL/F | apparent clearance of drug from eg, plasma |
| $C_{max}$ | maximum observed concentration |
| $CO_2$ | carbon dioxide (bicarbonate) |
| COVID-19 | coronavirus disease 2019 |
| CRF | case report form |
| CRO | contract research organization |
| CRU | clinical research unit |
| CSR | clinical study report |
| CT | clinical trial |
| CTMS | clinical trial management system |
| CYP | cytochrome P450 |

| Abbreviation | Term |
|--------------|-----------------------------------------|
| CYP3450 | cytochrome P450, family 3 |
| CYP3A | cytochrome P450, family 3, subfamily A |
| CYP3A4 | cytochrome P450 3A4 |
| CYP3A5 | cytochrome P450 3A5 |
| DILI | drug-induced liver injury |
| DMC | data monitoring committee |
| DNA | deoxyribonucleic acid |
| EC | ethics committee |
| ECC | emergency contact card |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDB | exposure during breastfeeding |
| EDP | exposure during pregnancy |
| EDR | extemporaneous dispensing record |
| eGFR | estimated glomerular filtration rate |
| EMA | European Medicines Agency |
| EU | European Union |
| EudraCT | European Clinical Trials Database |
| FIH | first in human |
| $f_{m}$ | fraction metabolized |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GLP | Good Laboratory Practice |
| HBcAb | hepatitis B core antibody |
| HBsAb | hepatitis B surface antibody |
| HBsAg | hepatitis B surface antigen |
| HCoV-229E | human coronavirus 229E |
| HCoV-HKU1 | human coronavirus HKU1 |
| HCoV-NL63 | human coronavirus NL63 |
| HCoV-OC43 | human coronavirus OC43 |
| HCV | hepatitis C virus |
| HCVAb | hepatitis C antibody |
| HIV | human immunodeficiency virus |
| HR | heart rate |
| HRT | hormone replacement therapy |
| IB | investigator's brochure |
| ICD | informed consent document |
| ICH | International Council for Harmonisation |
| ID | identification |
| IMP | investigational medicinal product |

| Abbreviation | Term |
|---|---|
| IND | investigational new drug |
| INR | international normalized ratio |
| IPAL | Investigational Product Accountability Log |
| IRB | institutional review board |
| IV | intravenous |
| kel | elimination rate constant |
| Ki | inhibition constant |
| LBBB | left bundle branch block |
| Loge | natural logarithm |
| LFT | liver function test |
| lnC <sub>max</sub> | log-transformed C <sub>max</sub> |
| lnAUC <sub>tau</sub> | log-transformed AUC <sub>tau</sub> |
| MAD | multiple ascending dose |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MERS | Middle East respiratory syndrome |
| msec | millisecond |
| N/A | not applicable |
| NHP | non-human primate |
| NOAEL | no-observed-adverse-effect level |
| NSAE | non-serious adverse event |
| NYHA | New York Heart Association |
| PCR | polymerase chain reaction |
| PCRU | Pfizer clinical research unit |
| PE | physical examination |
| рН | potential of hydrogen |
| PK | pharmacokinetic(s) |
| PR | pulse rate |
| PT | prothrombin time |
| PT-INR | prothrombin time-international normalized ratio |
| PVC | premature ventricular contraction/complex |
| q12h | every 12 hours |
| QD | once a day |
| QT | time from the beginning of the QRS complex to the end of the |
| | T wave |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |
| QTL | quality tolerance limit |
| qual | qualitative |
| RBC | red blood cell |

| Abbreviation | Term |
|------------------|-------------------------------------------------|
| RNA | ribonucleic acid |
| RR | respiratory rate |
| RT-PCR | reverse-transcriptase polymerase chain reaction |
| SAD | single ascending dose |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SARS-CoV-1 | severe acute respiratory syndrome coronavirus 1 |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SCr | serum creatinine |
| SmPC | Summary of product characteristics |
| SoA | schedule of activities |
| SOC | System Organ Class |
| SOP | standard operating procedure |
| SRSD | single reference safety document |
| SUSAR | suspected unexpected serious adverse reaction |
| t <sub>1/2</sub> | terminal half-life |
| T4 | thyroxine |
| TBili | total bilirubin |
| TEAE | treatment emergent adverse event |
| THC | tetrahydrocannabinol |
| $T_{\text{max}}$ | time to maximum concentration |
| TSH | thyroid stimulating hormone |
| ULN | upper limit of normal |
| US | United States |
| Vz/F | apparent volume of distribution |
| WBC | white blood cell |
| WHO | World Health Organization |
| WOCBP | woman/women of childbearing potential |

#### 11. REFERENCES

- IIsu A, Granneman G, Bertz R. Ritonavir: Clinical pharmacokinetics and interactions with other anti-HIV agents. Clin Pharmacokinet. 1998;35:275-91.
- WHO Situation Report 51. 11 March 2020 Available from: https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports. Accessed: 29 March 2020.
- Anand K, Ziebuhr J, Wadhwani P, et al. Coronavirus main proteinase (3CLpro) structure: basis for design of anti-SARS drugs. Science 2003;300:1763-7.
- <sup>4</sup> Ritonavir Single Reference Safety Document (SRSD): https://www.ema.europa.eu/en/documents/product-information/norvir-epar-product-information en.pdf
- Itraconazole Single Reference Safety Document (SRSD): SmPC Sporanox®, Belgium. https://www.janssen.com/belgium/sites/www\_janssen\_com\_belgium/files/prod\_files/live/mskp\_sporanoxdrank\_n.pdf
- Isoherranen N, Kunze KL, Allen KE, Nelson WL, Thummel KE. Role of itraconazole metabolites in CYP3A4 inhibition. Drug Metabolism and Disposition. 2004 Oct 1;32(10):1121-31.
- Liu L, Bello A, Dresser MJ, Heald D, Komjathy SF, O'Mara E, Rogge M, Stoch SA, Robertson SM. Best practices for the use of itraconazole as a replacement for ketoconazole in drug–drug interaction studies. The Journal of Clinical Pharmacology. 2016 Feb;56(2):143-51.